CLINICAL TRIAL: NCT05580003
Title: COVID-19: A MULTIPART, PHASE 1 STUDY WITH RANDOMIZED, DOUBLE-BLIND, SPONSOR-OPEN, PLACEBO-CONTROLLED, SINGLE- AND MULTIPLE-DOSE ESCALATION TO EVALUATE THE SAFETY, TOLERABILITY AND PHARMACOKINETICS OF PF-07817883 AND OPTIONAL OPEN-LABEL, RANDOMIZED STUDY TO EVALUATE RELATIVE BIOAVAILABILITY AND FOOD EFFECT OF SOLID ORAL FORMULATION AND OPTIONAL OPEN-LABEL, NON-RANDOMIZED STUDY TO EVALUATE METABOLISM AND EXCRETION OF PF-07817883 AND OPTIONAL RANDOMIZED, OPEN-LABEL STUDY TO ASSESS THE EFFECT OF PF-07817883 ON PHARMACOKINETICS OF MIDAZOLAM IN HEALTHY ADULT PARTICIPANTS
Brief Title: A Study to Learn Safety and Blood Levels of PF-07817883 in Healthy People
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: C5091001; 2022-002871-12 (EudraCT Number); 2022-002871-12 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-09

CONDITIONS: Healthy
Keywords: Oral Antiviral; COVID-19; Protease Inhibitor; Mpro; PF-07817883
MeSH Terms: conditions — COVID-19 | interventions — Midazolam; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: PART-1 and -2 are a randomized, double-blind, sponsor-open, placebo-controlled trial to evaluate safety, tolerability and PK of single and multiple escalating oral doses of PF 07817883 in healthy adult participants, respectively. PART-1 is crossover while PART-2 is parallel cohort study design. PART-2 of the study may also evaluate the safety, tolerability and PK in Japanese and Chinese participants. PART-3 is a randomized, open-label, cross-over, study to evaluate relative bioavailability and food effect of up to 2 new PF 07817883 oral formulations. PART-4 is an open label, non-randomized, single period cohort to evaluate the metabolism and excretion of PF 07817883. PART-5 is an open-label, randomized, cross-over cohort to evaluate the effect of steady state PF-07817883 on PK of midazolam in healthy participants. PART-6 is a sponsor-open, randomized, 3-treatment, 3-period, cross over study to evaluate safety, tolerability, and PK of PF 07817883 at supratherapeutic exposure.
Who Masked: Participant, Investigator
Masking Description: PART-1, 2 and 6 are double-blind, sponsor-open while PART-3, 4 and 5 are open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (25):
- PF-07817883 Dose 1 in PART-1 (Experimental)
  Interventions: Drug: PF-07817883
- PF-07817883 Dose 2 in PART-1 (Experimental)
  Interventions: Drug: PF-07817883
- PF-07817883 Dose 3 in PART-1 (Experimental)
  Interventions: Drug: PF-07817883
- PF-07817883 Dose 4 in PART-1 (Experimental)
  Interventions: Drug: PF-07817883
- PF-07817883 Dose 5 in PART-1 (Experimental): Optional dose levels
  Interventions: Drug: PF-07817883
- PF-07817883 Dose 6 in PART-1 (Experimental): Optional dose levels
  Interventions: Drug: PF-07817883
- Placebo in PART-1 (Placebo Comparator): A single dose of placebo
  Interventions: Drug: Placebo
- PF-07817883 DR1 in PART-2 (Experimental): DR=Dosing regimen; twice a day
  Interventions: Drug: PF-07817883
- PF-07817883 DR2 in PART-2 (Experimental)
  Interventions: Drug: PF-07817883
- PF-07817883 DR3 in PART-2 (Experimental): Optional dosing regimen
  Interventions: Drug: PF-07817883
- PF-07817883 DR4 in PART-2 (Experimental): Optional dosing regimen
  Interventions: Drug: PF-07817883
- PF-07817883 in Japanese in PART-2 (Experimental): Optional dosing regimen to be studied in Japanese population
  Interventions: Drug: PF-07817883
- PF-07817883 in Chinese in PART-2 (Experimental): Optional dosing regimen to be studied in Chinese population
  Interventions: Drug: PF-07817883
- Placebo in PART-2 (Placebo Comparator)
  Interventions: Drug: Placebo
- PF-07817883 Suspension Fasted in PART-3 (Experimental): PART-3 is optional
  Interventions: Drug: PF-07817883
- PF-07817883 FORM-1 Fasted in PART-3 (Experimental): First solid oral formulation (FORM1)
  Interventions: Drug: PF-07817883
- PF-07817883 FORM-2 Fasted in PART-3 (Experimental): Second solid oral formulations (FORM-2) is optional
  Interventions: Drug: PF-07817883
- PF-07817883 FORM-1 Fed in PART-3 (Experimental)
  Interventions: Drug: PF-07817883
- PF-07817883 FORM-2 Fed in PART-3 (Experimental)
  Interventions: Drug: PF-07817883
- PF-07817883 in PART-4 (Experimental): PART-4 is optional
  Interventions: Drug: PF-07817883
- Midazolam 5 mg in PART-5 (Experimental): Single dose of 5 mg alone
  Interventions: Drug: Midazolam
- Midazolam 5 mg with PF-07817883 in PART-5 (Experimental): Single dose of 5 mg on Day 10 with multiple doses (twice a day) of PF-07817883
  Interventions: Drug: PF-07817883; Drug: Midazolam
- PF-07817883 in PART-6 (Experimental): A single dose at supratherapeutic exposure administered as divided doses (1h apart)
  Interventions: Drug: PF-07817883
- Placebo in PART-6 (Placebo Comparator): A single dose of placebo administered as divided doses (1h apart)
  Interventions: Drug: Placebo
- Moxifloxacin 400 mg in PART-6 (open label) (Active Comparator): Moxifloxacin 400 mg at 0h followed by placebo at 1h
  Interventions: Drug: Placebo; Drug: Moxifloxacin

INTERVENTIONS:
Drug: PF-07817883 — Oral suspension or solid oral formulation(s)
  Arms: Midazolam 5 mg with PF-07817883 in PART-5; PF-07817883 DR1 in PART-2; PF-07817883 DR2 in PART-2; PF-07817883 DR3 in PART-2; PF-07817883 DR4 in PART-2; PF-07817883 Dose 1 in PART-1; PF-07817883 Dose 2 in PART-1; PF-07817883 Dose 3 in PART-1; PF-07817883 Dose 4 in PART-1; PF-07817883 Dose 5 in PART-1; PF-07817883 Dose 6 in PART-1; PF-07817883 FORM-1 Fasted in PART-3; PF-07817883 FORM-1 Fed in PART-3; PF-07817883 FORM-2 Fasted in PART-3; PF-07817883 FORM-2 Fed in PART-3; PF-07817883 Suspension Fasted in PART-3; PF-07817883 in Chinese in PART-2; PF-07817883 in Japanese in PART-2; PF-07817883 in PART-4; PF-07817883 in PART-6
Drug: Placebo — Placebo suspension
  Arms: Moxifloxacin 400 mg in PART-6 (open label); Placebo in PART-1; Placebo in PART-2; Placebo in PART-6
Drug: Midazolam — midazolam oral solution
  Arms: Midazolam 5 mg in PART-5; Midazolam 5 mg with PF-07817883 in PART-5
Drug: Moxifloxacin — Moxifloxacin 400 mg tablet
  Arms: Moxifloxacin 400 mg in PART-6 (open label)

SUMMARY:
The purpose of this clinical trial is to learn if the study medicine (called PF-07817883) is safe and how it goes in and out of the body in healthy people. PF-07817883 is for the potential treatment of COVID-19. Participants will take PF-07817883 by mouth up to 2 times a day. This study may also evaluate how much PF-07817883 gets into the body when taken as pill. We may study if people's diets can affect this study medicine. We may also examine how PF-07817883 is processed and removed by the human body. Finally, we may look into if PF-07817883 has potential to interact with midazolam.

DETAILED DESCRIPTION:
Combined 6-part study. Part-1: Single Ascending dose Part-2: Multiple Ascending Dose Part-3: Relative bioavailability and food effect Part-4: Metabolism and Excretion Part-5: Drug-drug interaction with midazolam Part-6: Supratherapeutic exposure Part-1,2 and 6 are double blind, sponsor open and Part-3,4 and 5 are open label study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects between ages of 18-60 years. Male only in part-4.
* Body Mass Index (BMI) of 17.5 to 30.5kg/m2; and a total body weight >50kg (110lbs). A body weight of >45 kg may be considered in selected cases.
* Japanese subjects who have four Japanese biologic grandparents born in Japan
* Chinese participants who were born in mainland China and both parents are of the Chinese descent.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing)
* Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy, intestinal resection).
* Positive test result for SARS-CoV-2 infection at the time of screening or Day-1.
* Have received COVID-19 vaccine within 7 days before screening or have received only one of the 2 required doses of COVID-19 vaccine
* Use of tobacco or nicotine containing products in excess of the equivalents of 5 cigarettes per day or 2 chews of tobacco per day
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 28 days or 5 half lives (whichever is longer) prior to the first dose of study intervention.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- New Haven Clinical Research Unit, New Haven, Connecticut, United States
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5091001

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 94 participants were enrolled across Belgium and United States.
Groups:
- P1: C1: Placebo,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg, Fast: In this cohort (C), participants received a single dose of placebo as an oral suspension in the fasted (fast) state on Day 1 of Period 1 followed by a single dose of PF-07817883 1500 milligram (mg) as an oral suspension in the fasted state on Day 1 of Period 2. Participants were administered a single dose of PF-07817883 4000 mg as an oral suspension in the fasted state on Day 1 of Period 3. There was a washout of at least 5 days between two doses.
- P1: C1: PF-07817883 150mg,Fast/Placebo,Fast/PF-07817883 4000mg,Fast: Participants received a single dose of PF-07817883 150 mg as an oral suspension in the fasted state on Day 1 of Period 1 followed by a single dose of placebo as an oral suspension in the fasted state on Day 1 of Period 2. Participants were administered a single dose of PF-07817883 4000 mg as an oral suspension in the fasted state on Day 1 of Period 3. There was a washout of at least 5 days between two doses.
- P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/Placebo,Fast: Participants received a single dose of PF-07817883 150 mg as an oral suspension in the fasted state on Day 1 of Period 1 followed by a single dose of PF-07817883 1500 mg as an oral suspension in the fasted state on Day 1 of Period 2. Participants were administered a single dose of placebo as an oral suspension in the fasted state on Day 1 of Period 3. There was a washout of at least 5 days between two doses.
- P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg,Fast: Participants received a single dose of PF-07817883 150 mg as an oral suspension in the fasted state on Day 1 of Period 1 followed by a single dose of PF-07817883 1500 mg as an oral suspension in the fasted state on Day 1 of Period 2. Participants were administered a single dose of PF-07817883 4000 mg as an oral suspension in the fasted state on Day 1 of Period 3. There was a washout of at least 5 days between two doses.
- P1: C2: Placebo,Fast/PF-07817883 3000mg,Fast/Placebo,Fed: Participants received a single dose of placebo as an oral suspension in the fasted state on Day 1 of Period 1 followed by a single dose of PF-07817883 3000 mg as an oral suspension in the fasted state on Day 1 of Period 2. Participants were administered a single dose of placebo as an oral suspension in the fed state on Day 1 of Period 3. There was a washout of at least 5 days between two doses.
- P1: C2: PF-07817883 500mg,Fast/Placebo,Fast/PF-07817883 500mg,Fed: Participants received a single dose of PF-07817883 500 mg as an oral suspension in the fasted state on Day 1 of Period 1 followed by a single dose of placebo as an oral suspension in the fasted state on Day 1 of Period 2. Participants were administered a single dose of PF-07817883 500 mg as an oral suspension in the fed state on Day 1 of Period 3. There was a washout of at least 5 days between two doses.
- P1: C2: PF-07817883 500mg,Fast/PF-07817883 3000mg,Fast/PF-07817883 500mg,Fed: Participants received a single dose of PF-07817883 500 mg as an oral suspension in the fasted state on Day 1 of Period 1 followed by a single dose of PF-07817883 3000 mg as an oral suspension in the fasted state on Day 1 of Period 2. Participants were administered a single dose of PF-07817883 500 mg as an oral suspension in the fed state on Day 1 of Period 3. There was a washout of at least 5 days between two doses.
- Part 2: Placebo (Suspension) BID, Fasted: Participants received placebo oral suspension twice a day (BID) administered every 12 hours on Days 1 to 9. On Day 10, participants received only one dose of placebo in the morning under fasted conditions.
- Part 2: PF-07817883 200 mg (Suspension) BID, Fasted: Participants received PF-07817883 200 mg oral suspension BID administered every 12 hours on Days 1 to 9. On Day 10, participants received only one dose of PF-07817883 200 mg in the morning under fasted conditions.
- Part 2: PF-07817883 600 mg (Suspension) BID, Fasted: Participants received PF-07817883 600 mg oral suspension BID administered every 12 hours on Days 1 to 9. On Day 10, participants received only one dose of PF-07817883 600 mg in the morning under fasted conditions.
- Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted: Participants received PF-07817883 1500 mg oral suspension BID administered every 12 hours on Days 1 to 9. On Day 10, participants received only one dose of PF-07817883 1500 mg in the morning under fasted conditions.
- Part 2: Placebo (Suspension) BID, Fasted, Chinese: Chinese participants received placebo oral suspension BID administered every 12 hours on Days 1 to 9. On Day 10, participants received only one dose of placebo in the morning under fasted conditions.
- Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese: Chinese participants received PF-07817883 600 mg oral suspension BID administered every 12 hours on Days 1 to 9. On Day 10, participants received only one dose of PF-07817883 600 mg in the morning under fasted conditions.
- Part 3: Treatment Sequence ABCD: Participants received treatments A, B, C and D in Period 1, 2, 3 and 4 respectively. Treatment A: Single dose of PF-07817883 spray dried dispersion (SDD) 600 mg tablets in fasted conditions. Treatment B: Single dose of PF-07817883 crystalline 600 mg tablet in fasted conditions. Treatment C: Single dose of PF-07817883 600 mg suspension in fasted conditions. Treatment D: Single dose of PF-07817883 SDD 600 mg tablet in fed conditions. There was a washout of at least 3 days between 2 doses.
- Part 3: Treatment Sequence BCAD: Participants received treatments B, C, A and D in Period 1, 2, 3 and 4 respectively. Treatment B: Single dose of PF-07817883 crystalline 600 mg tablet in fasted conditions. Treatment C: Single dose of PF-07817883 600 mg suspension in fasted conditions. Treatment A: Single dose of PF-07817883 SDD 600 mg tablets in fasted conditions. Treatment D: Single dose of PF-07817883 SDD 600 mg tablet in fed conditions. There was a washout of at least 3 days between 2 doses.
- Part 3: Treatment Sequence CABD: Participants received treatments C, A, B and D in Period 1, 2, 3 and 4 respectively. Treatment C: Single dose of PF-07817883 600 mg suspension in fasted conditions. Treatment A: Single dose of PF-07817883 SDD 600 mg tablets in fasted conditions. Treatment B: Single dose of PF-07817883 crystalline 600 mg tablet in fasted conditions. Treatment D: Single dose of PF-07817883 SDD 600 mg tablet in fed conditions. There was a washout of at least 3 days between 2 doses.
- Part 3: Treatment Sequence BACE: Participants received treatments B, A, C and E in Period 1, 2, 3 and 4 respectively. Treatment B: Single dose of PF-07817883 crystalline 600 mg tablet in fasted conditions. Treatment A: Single dose of PF-07817883 SDD 600 mg tablets in fasted conditions. Treatment C: Single dose of PF-07817883 600 mg suspension in fasted conditions. Treatment E: Single dose of PF-07817883 crystalline 600 mg tablet in fed conditions. There was a washout of at least 3 days between 2 doses.
- Part 3: Treatment Sequence ACBE: Participants received treatments A, C, B and E in Period 1, 2, 3 and 4 respectively. Treatment A: Single dose of PF-07817883 SDD 600 mg tablets in fasted conditions. Treatment C: Single dose of PF-07817883 600 mg suspension in fasted conditions. Treatment B: Single dose of PF-07817883 crystalline 600 mg tablet in fasted conditions. Treatment E: Single dose of PF-07817883 crystalline 600 mg tablet in fed conditions. There was a washout of at least 3 days between 2 doses.
- Part 3: Treatment Sequence CBAE: Participants received treatments C, B, A and E in Period 1, 2, 3 and 4 respectively. Treatment C: Single dose of PF-07817883 600 mg suspension in fasted conditions. Treatment B: Single dose of PF-07817883 crystalline 600 mg tablet in fasted conditions. Treatment A: Single dose of PF-07817883 SDD 600 mg tablets in fasted conditions. Treatment E: Single dose of PF-07817883 crystalline 600 mg tablet in fed conditions. There was a washout of at least 3 days between 2 doses.
- Part 4: PF-07817883 600 mg (Suspension), Fasted: Participants received a single dose of PF-07817883 600 mg oral suspension on Day 1 following an overnight fast of approximately 10 hours.
- Part 5: Treatment Sequence AB: Participants received a single dose of midazolam 5 mg orally on Day 1 of Period 1 followed by a 2-day washout period. In Period 2, participants received PF-07817883 BID orally for 10 days followed by single dose of midazolam 5 mg on Day 10 followed by a washout of at least 7 days.
- Part 5: Treatment Sequence BA: In Period 1, participants received PF-07817883 BID orally for 10 days and on Day 10, participants received a single oral dose of 5 mg midazolam administered with PF-07817883 followed by a washout of at least 7 days. In Period 2, participants received a single dose of midazolam 5 mg orally followed by a 2-day washout period.
- Part 6: Treatment Sequence ABC: Participants received treatment A, B and C in Period 1, 2 and 3 respectively. Treatment A: PF-07817883 6000 mg oral suspension administered as 2 split doses of 3000 mg at 0 and 1 hour under fasted conditions. Treatment B: Single dose of Placebo oral suspension following an overnight fast of at least 10 hours. Treatment C: Single dose of Moxifloxacin 400 mg oral tablet at 0 hour and placebo at 1 hour following an overnight fast of at least 10 hours. Each period was separated by a washout of at least 7 days.
- Part 6: Treatment Sequence BCA: Participants received treatment B, C and A in Period 1, 2 and 3 respectively. Treatment B: Single dose of Placebo oral suspension following an overnight fast of at least 10 hours. Treatment C: Single dose of Moxifloxacin 400 mg oral tablet at 0 hour and placebo at 1 hour following an overnight fast of at least 10 hours. Treatment A: PF-07817883 6000 mg oral suspension administered as 2 split doses of 3000 mg at 0 and 1 hour under fasted conditions. Each period was separated by a washout of at least 7 days.
- Part 6: Treatment Sequence CAB: Participants received treatment C, A and B in Period 1, 2 and 3 respectively. Treatment C: Single dose of Moxifloxacin 400 mg oral tablet at 0 hour and placebo at 1 hour following an overnight fast of at least 10 hours. Treatment A: PF-07817883 6000 mg oral suspension administered as 2 split doses of 3000 mg at 0 and 1 hour under fasted conditions. Treatment B: Single dose of Placebo oral suspension following an overnight fast of at least 10 hours. Each period was separated by a washout of at least 7 days.
- Part 6: Treatment Sequence BAC: Participants received treatment B, A and C in Period 1, 2 and 3 respectively. Treatment B: Single dose of Placebo oral suspension following an overnight fast of at least 10 hours. Treatment A: PF-07817883 6000 mg oral suspension administered as 2 split doses of 3000 mg at 0 and 1 hour under fasted conditions. Treatment C: Single dose of Moxifloxacin 400 mg oral tablet at 0 hour and placebo at 1 hour following an overnight fast of at least 10 hours. Each period was separated by a washout of at least 7 days.
- Part 6: Treatment Sequence ACB: Participants received treatment A, C and B in Period 1, 2 and 3 respectively. Treatment A: PF-07817883 6000 mg oral suspension administered as 2 split doses of 3000 mg at 0 and 1 hour under fasted conditions. Treatment C: Single dose of Moxifloxacin 400 mg oral tablet at 0 hour and placebo at 1 hour following an overnight fast of at least 10 hours. Treatment B: Single dose of Placebo oral suspension following an overnight fast of at least 10 hours. Each period was separated by a washout of at least 7 days.
- Part 6: Treatment Sequence CBA: Participants received treatment C, B and A in Period 1, 2 and 3 respectively. Treatment C: Single dose of Moxifloxacin 400 mg oral tablet at 0 hour and placebo at 1 hour following an overnight fast of at least 10 hours. Treatment B: Single dose of Placebo oral suspension following an overnight fast of at least 10 hours. Treatment A: PF-07817883 6000 mg oral suspension administered as 2 split doses of 3000 mg at 0 and 1 hour under fasted conditions. Each period was separated by a washout of at least 7 days.
Period: Part (P) 1 Treatment Period 1 (Day 1)
Arm/Group | P1: C1: Placebo,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg, Fast | P1: C1: PF-07817883 150mg,Fast/Placebo,Fast/PF-07817883 4000mg,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/Placebo,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg,Fast | P1: C2: Placebo,Fast/PF-07817883 3000mg,Fast/Placebo,Fed | P1: C2: PF-07817883 500mg,Fast/Placebo,Fast/PF-07817883 500mg,Fed | P1: C2: PF-07817883 500mg,Fast/PF-07817883 3000mg,Fast/PF-07817883 500mg,Fed | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese | Part 3: Treatment Sequence ABCD | Part 3: Treatment Sequence BCAD | Part 3: Treatment Sequence CABD | Part 3: Treatment Sequence BACE | Part 3: Treatment Sequence ACBE | Part 3: Treatment Sequence CBAE | Part 4: PF-07817883 600 mg (Suspension), Fasted | Part 5: Treatment Sequence AB | Part 5: Treatment Sequence BA | Part 6: Treatment Sequence ABC | Part 6: Treatment Sequence BCA | Part 6: Treatment Sequence CAB | Part 6: Treatment Sequence BAC | Part 6: Treatment Sequence ACB | Part 6: Treatment Sequence CBA
Started | 2 | 2 | 2 | 2 | 2 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1: Washout 1 (up to 5 Days)
Arm/Group | P1: C1: Placebo,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg, Fast | P1: C1: PF-07817883 150mg,Fast/Placebo,Fast/PF-07817883 4000mg,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/Placebo,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg,Fast | P1: C2: Placebo,Fast/PF-07817883 3000mg,Fast/Placebo,Fed | P1: C2: PF-07817883 500mg,Fast/Placebo,Fast/PF-07817883 500mg,Fed | P1: C2: PF-07817883 500mg,Fast/PF-07817883 3000mg,Fast/PF-07817883 500mg,Fed | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese | Part 3: Treatment Sequence ABCD | Part 3: Treatment Sequence BCAD | Part 3: Treatment Sequence CABD | Part 3: Treatment Sequence BACE | Part 3: Treatment Sequence ACBE | Part 3: Treatment Sequence CBAE | Part 4: PF-07817883 600 mg (Suspension), Fasted | Part 5: Treatment Sequence AB | Part 5: Treatment Sequence BA | Part 6: Treatment Sequence ABC | Part 6: Treatment Sequence BCA | Part 6: Treatment Sequence CAB | Part 6: Treatment Sequence BAC | Part 6: Treatment Sequence ACB | Part 6: Treatment Sequence CBA
Started | 2 (Participants who started washout 1 of Part 1.) | 2 (Participants who started washout 1 of Part 1.) | 2 (Participants who started washout 1 of Part 1.) | 2 (Participants who started washout 1 of Part 1.) | 2 (Participants who started washout 1 of Part 1.) | 2 (Participants who started washout 1 of Part 1.) | 3 (Participants who started washout 1 of Part 1.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 2 | 2 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1 Treatment Period 2 (Day 1)
Arm/Group | P1: C1: Placebo,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg, Fast | P1: C1: PF-07817883 150mg,Fast/Placebo,Fast/PF-07817883 4000mg,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/Placebo,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg,Fast | P1: C2: Placebo,Fast/PF-07817883 3000mg,Fast/Placebo,Fed | P1: C2: PF-07817883 500mg,Fast/Placebo,Fast/PF-07817883 500mg,Fed | P1: C2: PF-07817883 500mg,Fast/PF-07817883 3000mg,Fast/PF-07817883 500mg,Fed | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese | Part 3: Treatment Sequence ABCD | Part 3: Treatment Sequence BCAD | Part 3: Treatment Sequence CABD | Part 3: Treatment Sequence BACE | Part 3: Treatment Sequence ACBE | Part 3: Treatment Sequence CBAE | Part 4: PF-07817883 600 mg (Suspension), Fasted | Part 5: Treatment Sequence AB | Part 5: Treatment Sequence BA | Part 6: Treatment Sequence ABC | Part 6: Treatment Sequence BCA | Part 6: Treatment Sequence CAB | Part 6: Treatment Sequence BAC | Part 6: Treatment Sequence ACB | Part 6: Treatment Sequence CBA
Started | 2 (Participants who started Period 2 of Part 1.) | 2 (Participants who started Period 2 of Part 1.) | 2 (Participants who started Period 2 of Part 1.) | 2 (Participants who started Period 2 of Part 1.) | 2 (Participants who started Period 2 of Part 1.) | 2 (Participants who started Period 2 of Part 1.) | 3 (Participants who started Period 2 of Part 1.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 1 | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1: Washout 2 (up to 5 Days)
Arm/Group | P1: C1: Placebo,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg, Fast | P1: C1: PF-07817883 150mg,Fast/Placebo,Fast/PF-07817883 4000mg,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/Placebo,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg,Fast | P1: C2: Placebo,Fast/PF-07817883 3000mg,Fast/Placebo,Fed | P1: C2: PF-07817883 500mg,Fast/Placebo,Fast/PF-07817883 500mg,Fed | P1: C2: PF-07817883 500mg,Fast/PF-07817883 3000mg,Fast/PF-07817883 500mg,Fed | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese | Part 3: Treatment Sequence ABCD | Part 3: Treatment Sequence BCAD | Part 3: Treatment Sequence CABD | Part 3: Treatment Sequence BACE | Part 3: Treatment Sequence ACBE | Part 3: Treatment Sequence CBAE | Part 4: PF-07817883 600 mg (Suspension), Fasted | Part 5: Treatment Sequence AB | Part 5: Treatment Sequence BA | Part 6: Treatment Sequence ABC | Part 6: Treatment Sequence BCA | Part 6: Treatment Sequence CAB | Part 6: Treatment Sequence BAC | Part 6: Treatment Sequence ACB | Part 6: Treatment Sequence CBA
Started | 2 (Participants who started washout 2 of Part 1.) | 2 (Participants who started washout 2 of Part 1.) | 2 (Participants who started washout 2 of Part 1.) | 1 (Participants who started washout 2 of Part 1.) | 2 (Participants who started washout 2 of Part 1.) | 1 (Participants who started washout 2 of Part 1.) | 3 (Participants who started washout 2 of Part 1.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 2 | 2 | 1 | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 1: Treatment Period 3 (Day 1)
Arm/Group | P1: C1: Placebo,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg, Fast | P1: C1: PF-07817883 150mg,Fast/Placebo,Fast/PF-07817883 4000mg,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/Placebo,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg,Fast | P1: C2: Placebo,Fast/PF-07817883 3000mg,Fast/Placebo,Fed | P1: C2: PF-07817883 500mg,Fast/Placebo,Fast/PF-07817883 500mg,Fed | P1: C2: PF-07817883 500mg,Fast/PF-07817883 3000mg,Fast/PF-07817883 500mg,Fed | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese | Part 3: Treatment Sequence ABCD | Part 3: Treatment Sequence BCAD | Part 3: Treatment Sequence CABD | Part 3: Treatment Sequence BACE | Part 3: Treatment Sequence ACBE | Part 3: Treatment Sequence CBAE | Part 4: PF-07817883 600 mg (Suspension), Fasted | Part 5: Treatment Sequence AB | Part 5: Treatment Sequence BA | Part 6: Treatment Sequence ABC | Part 6: Treatment Sequence BCA | Part 6: Treatment Sequence CAB | Part 6: Treatment Sequence BAC | Part 6: Treatment Sequence ACB | Part 6: Treatment Sequence CBA
Started | 2 (Participants who started Period 3 of Part 1.) | 2 (Participants who started Period 3 of Part 1.) | 2 (Participants who started Period 3 of Part 1.) | 1 (Participants who started Period 3 of Part 1.) | 2 (Participants who started Period 3 of Part 1.) | 1 (Participants who started Period 3 of Part 1.) | 3 (Participants who started Period 3 of Part 1.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 1 | 2 | 1 | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2 (up to 10 Days)
Arm/Group | P1: C1: Placebo,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg, Fast | P1: C1: PF-07817883 150mg,Fast/Placebo,Fast/PF-07817883 4000mg,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/Placebo,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg,Fast | P1: C2: Placebo,Fast/PF-07817883 3000mg,Fast/Placebo,Fed | P1: C2: PF-07817883 500mg,Fast/Placebo,Fast/PF-07817883 500mg,Fed | P1: C2: PF-07817883 500mg,Fast/PF-07817883 3000mg,Fast/PF-07817883 500mg,Fed | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese | Part 3: Treatment Sequence ABCD | Part 3: Treatment Sequence BCAD | Part 3: Treatment Sequence CABD | Part 3: Treatment Sequence BACE | Part 3: Treatment Sequence ACBE | Part 3: Treatment Sequence CBAE | Part 4: PF-07817883 600 mg (Suspension), Fasted | Part 5: Treatment Sequence AB | Part 5: Treatment Sequence BA | Part 6: Treatment Sequence ABC | Part 6: Treatment Sequence BCA | Part 6: Treatment Sequence CAB | Part 6: Treatment Sequence BAC | Part 6: Treatment Sequence ACB | Part 6: Treatment Sequence CBA
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 (Participants enrolled in Part 2 of the study.) | 4 (Participants enrolled in Part 2 of the study.) | 4 (Participants enrolled in Part 2 of the study.) | 4 (Participants enrolled in Part 2 of the study.) | 1 (Participants enrolled in Part 2 of the study.) | 3 (Participants enrolled in Part 2 of the study.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 4 | 3 | 4 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3 Period 1 (Day 1)
Arm/Group | P1: C1: Placebo,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg, Fast | P1: C1: PF-07817883 150mg,Fast/Placebo,Fast/PF-07817883 4000mg,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/Placebo,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg,Fast | P1: C2: Placebo,Fast/PF-07817883 3000mg,Fast/Placebo,Fed | P1: C2: PF-07817883 500mg,Fast/Placebo,Fast/PF-07817883 500mg,Fed | P1: C2: PF-07817883 500mg,Fast/PF-07817883 3000mg,Fast/PF-07817883 500mg,Fed | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese | Part 3: Treatment Sequence ABCD | Part 3: Treatment Sequence BCAD | Part 3: Treatment Sequence CABD | Part 3: Treatment Sequence BACE | Part 3: Treatment Sequence ACBE | Part 3: Treatment Sequence CBAE | Part 4: PF-07817883 600 mg (Suspension), Fasted | Part 5: Treatment Sequence AB | Part 5: Treatment Sequence BA | Part 6: Treatment Sequence ABC | Part 6: Treatment Sequence BCA | Part 6: Treatment Sequence CAB | Part 6: Treatment Sequence BAC | Part 6: Treatment Sequence ACB | Part 6: Treatment Sequence CBA
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (Participants enrolled in Part 3 of the study.) | 2 (Participants enrolled in Part 3 of the study.) | 2 (Participants enrolled in Part 3 of the study.) | 2 (Participants enrolled in Part 3 of the study.) | 2 (Participants enrolled in Part 3 of the study.) | 2 (Participants enrolled in Part 3 of the study.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3: Washout 1 (up to 3 Days)
Arm/Group | P1: C1: Placebo,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg, Fast | P1: C1: PF-07817883 150mg,Fast/Placebo,Fast/PF-07817883 4000mg,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/Placebo,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg,Fast | P1: C2: Placebo,Fast/PF-07817883 3000mg,Fast/Placebo,Fed | P1: C2: PF-07817883 500mg,Fast/Placebo,Fast/PF-07817883 500mg,Fed | P1: C2: PF-07817883 500mg,Fast/PF-07817883 3000mg,Fast/PF-07817883 500mg,Fed | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese | Part 3: Treatment Sequence ABCD | Part 3: Treatment Sequence BCAD | Part 3: Treatment Sequence CABD | Part 3: Treatment Sequence BACE | Part 3: Treatment Sequence ACBE | Part 3: Treatment Sequence CBAE | Part 4: PF-07817883 600 mg (Suspension), Fasted | Part 5: Treatment Sequence AB | Part 5: Treatment Sequence BA | Part 6: Treatment Sequence ABC | Part 6: Treatment Sequence BCA | Part 6: Treatment Sequence CAB | Part 6: Treatment Sequence BAC | Part 6: Treatment Sequence ACB | Part 6: Treatment Sequence CBA
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (Participants who started washout 1 of Part 3.) | 2 (Participants who started washout 1 of Part 3.) | 2 (Participants who started washout 1 of Part 3.) | 2 (Participants who started washout 1 of Part 3.) | 2 (Participants who started washout 1 of Part 3.) | 2 (Participants who started washout 1 of Part 3.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3: Period 2 (Day 1)
Arm/Group | P1: C1: Placebo,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg, Fast | P1: C1: PF-07817883 150mg,Fast/Placebo,Fast/PF-07817883 4000mg,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/Placebo,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg,Fast | P1: C2: Placebo,Fast/PF-07817883 3000mg,Fast/Placebo,Fed | P1: C2: PF-07817883 500mg,Fast/Placebo,Fast/PF-07817883 500mg,Fed | P1: C2: PF-07817883 500mg,Fast/PF-07817883 3000mg,Fast/PF-07817883 500mg,Fed | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese | Part 3: Treatment Sequence ABCD | Part 3: Treatment Sequence BCAD | Part 3: Treatment Sequence CABD | Part 3: Treatment Sequence BACE | Part 3: Treatment Sequence ACBE | Part 3: Treatment Sequence CBAE | Part 4: PF-07817883 600 mg (Suspension), Fasted | Part 5: Treatment Sequence AB | Part 5: Treatment Sequence BA | Part 6: Treatment Sequence ABC | Part 6: Treatment Sequence BCA | Part 6: Treatment Sequence CAB | Part 6: Treatment Sequence BAC | Part 6: Treatment Sequence ACB | Part 6: Treatment Sequence CBA
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (Participants who started Period 2 of Part 3.) | 2 (Participants who started Period 2 of Part 3.) | 2 (Participants who started Period 2 of Part 3.) | 2 (Participants who started Period 2 of Part 3.) | 2 (Participants who started Period 2 of Part 3.) | 2 (Participants who started Period 2 of Part 3.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3: Washout 2 (up to 3 Days)
Arm/Group | P1: C1: Placebo,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg, Fast | P1: C1: PF-07817883 150mg,Fast/Placebo,Fast/PF-07817883 4000mg,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/Placebo,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg,Fast | P1: C2: Placebo,Fast/PF-07817883 3000mg,Fast/Placebo,Fed | P1: C2: PF-07817883 500mg,Fast/Placebo,Fast/PF-07817883 500mg,Fed | P1: C2: PF-07817883 500mg,Fast/PF-07817883 3000mg,Fast/PF-07817883 500mg,Fed | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese | Part 3: Treatment Sequence ABCD | Part 3: Treatment Sequence BCAD | Part 3: Treatment Sequence CABD | Part 3: Treatment Sequence BACE | Part 3: Treatment Sequence ACBE | Part 3: Treatment Sequence CBAE | Part 4: PF-07817883 600 mg (Suspension), Fasted | Part 5: Treatment Sequence AB | Part 5: Treatment Sequence BA | Part 6: Treatment Sequence ABC | Part 6: Treatment Sequence BCA | Part 6: Treatment Sequence CAB | Part 6: Treatment Sequence BAC | Part 6: Treatment Sequence ACB | Part 6: Treatment Sequence CBA
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (Participants who started washout 2 of Part 3.) | 2 (Participants who started washout 2 of Part 3.) | 2 (Participants who started washout 2 of Part 3.) | 2 (Participants who started washout 2 of Part 3.) | 2 (Participants who started washout 2 of Part 3.) | 2 (Participants who started washout 2 of Part 3.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3: Period 3 (Day 1)
Arm/Group | P1: C1: Placebo,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg, Fast | P1: C1: PF-07817883 150mg,Fast/Placebo,Fast/PF-07817883 4000mg,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/Placebo,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg,Fast | P1: C2: Placebo,Fast/PF-07817883 3000mg,Fast/Placebo,Fed | P1: C2: PF-07817883 500mg,Fast/Placebo,Fast/PF-07817883 500mg,Fed | P1: C2: PF-07817883 500mg,Fast/PF-07817883 3000mg,Fast/PF-07817883 500mg,Fed | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese | Part 3: Treatment Sequence ABCD | Part 3: Treatment Sequence BCAD | Part 3: Treatment Sequence CABD | Part 3: Treatment Sequence BACE | Part 3: Treatment Sequence ACBE | Part 3: Treatment Sequence CBAE | Part 4: PF-07817883 600 mg (Suspension), Fasted | Part 5: Treatment Sequence AB | Part 5: Treatment Sequence BA | Part 6: Treatment Sequence ABC | Part 6: Treatment Sequence BCA | Part 6: Treatment Sequence CAB | Part 6: Treatment Sequence BAC | Part 6: Treatment Sequence ACB | Part 6: Treatment Sequence CBA
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (Participants who started Period 3 of Part 3.) | 2 (Participants who started Period 3 of Part 3.) | 2 (Participants who started Period 3 of Part 3.) | 2 (Participants who started Period 3 of Part 3.) | 2 (Participants who started Period 3 of Part 3.) | 2 (Participants who started Period 3 of Part 3.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3: Washout 3 (up to 3 Days)
Arm/Group | P1: C1: Placebo,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg, Fast | P1: C1: PF-07817883 150mg,Fast/Placebo,Fast/PF-07817883 4000mg,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/Placebo,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg,Fast | P1: C2: Placebo,Fast/PF-07817883 3000mg,Fast/Placebo,Fed | P1: C2: PF-07817883 500mg,Fast/Placebo,Fast/PF-07817883 500mg,Fed | P1: C2: PF-07817883 500mg,Fast/PF-07817883 3000mg,Fast/PF-07817883 500mg,Fed | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese | Part 3: Treatment Sequence ABCD | Part 3: Treatment Sequence BCAD | Part 3: Treatment Sequence CABD | Part 3: Treatment Sequence BACE | Part 3: Treatment Sequence ACBE | Part 3: Treatment Sequence CBAE | Part 4: PF-07817883 600 mg (Suspension), Fasted | Part 5: Treatment Sequence AB | Part 5: Treatment Sequence BA | Part 6: Treatment Sequence ABC | Part 6: Treatment Sequence BCA | Part 6: Treatment Sequence CAB | Part 6: Treatment Sequence BAC | Part 6: Treatment Sequence ACB | Part 6: Treatment Sequence CBA
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (Participants who started washout 3 of Part 3.) | 2 (Participants who started washout 3 of Part 3.) | 2 (Participants who started washout 3 of Part 3.) | 2 (Participants who started washout 3 of Part 3.) | 2 (Participants who started washout 3 of Part 3.) | 2 (Participants who started washout 3 of Part 3.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 3: Period 4 (Day 1)
Arm/Group | P1: C1: Placebo,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg, Fast | P1: C1: PF-07817883 150mg,Fast/Placebo,Fast/PF-07817883 4000mg,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/Placebo,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg,Fast | P1: C2: Placebo,Fast/PF-07817883 3000mg,Fast/Placebo,Fed | P1: C2: PF-07817883 500mg,Fast/Placebo,Fast/PF-07817883 500mg,Fed | P1: C2: PF-07817883 500mg,Fast/PF-07817883 3000mg,Fast/PF-07817883 500mg,Fed | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese | Part 3: Treatment Sequence ABCD | Part 3: Treatment Sequence BCAD | Part 3: Treatment Sequence CABD | Part 3: Treatment Sequence BACE | Part 3: Treatment Sequence ACBE | Part 3: Treatment Sequence CBAE | Part 4: PF-07817883 600 mg (Suspension), Fasted | Part 5: Treatment Sequence AB | Part 5: Treatment Sequence BA | Part 6: Treatment Sequence ABC | Part 6: Treatment Sequence BCA | Part 6: Treatment Sequence CAB | Part 6: Treatment Sequence BAC | Part 6: Treatment Sequence ACB | Part 6: Treatment Sequence CBA
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 (Participants who started Period 4 of Part 3.) | 2 (Participants who started Period 4 of Part 3.) | 2 (Participants who started Period 4 of Part 3.) | 2 (Participants who started Period 4 of Part 3.) | 2 (Participants who started Period 4 of Part 3.) | 2 (Participants who started Period 4 of Part 3.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 4 (Day 1 to Day 11)
Arm/Group | P1: C1: Placebo,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg, Fast | P1: C1: PF-07817883 150mg,Fast/Placebo,Fast/PF-07817883 4000mg,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/Placebo,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg,Fast | P1: C2: Placebo,Fast/PF-07817883 3000mg,Fast/Placebo,Fed | P1: C2: PF-07817883 500mg,Fast/Placebo,Fast/PF-07817883 500mg,Fed | P1: C2: PF-07817883 500mg,Fast/PF-07817883 3000mg,Fast/PF-07817883 500mg,Fed | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese | Part 3: Treatment Sequence ABCD | Part 3: Treatment Sequence BCAD | Part 3: Treatment Sequence CABD | Part 3: Treatment Sequence BACE | Part 3: Treatment Sequence ACBE | Part 3: Treatment Sequence CBAE | Part 4: PF-07817883 600 mg (Suspension), Fasted | Part 5: Treatment Sequence AB | Part 5: Treatment Sequence BA | Part 6: Treatment Sequence ABC | Part 6: Treatment Sequence BCA | Part 6: Treatment Sequence CAB | Part 6: Treatment Sequence BAC | Part 6: Treatment Sequence ACB | Part 6: Treatment Sequence CBA
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 (Participants enrolled in Part 4 of the study.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 5: Sequence AB: Period 1 (Day 1)
Arm/Group | P1: C1: Placebo,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg, Fast | P1: C1: PF-07817883 150mg,Fast/Placebo,Fast/PF-07817883 4000mg,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/Placebo,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg,Fast | P1: C2: Placebo,Fast/PF-07817883 3000mg,Fast/Placebo,Fed | P1: C2: PF-07817883 500mg,Fast/Placebo,Fast/PF-07817883 500mg,Fed | P1: C2: PF-07817883 500mg,Fast/PF-07817883 3000mg,Fast/PF-07817883 500mg,Fed | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese | Part 3: Treatment Sequence ABCD | Part 3: Treatment Sequence BCAD | Part 3: Treatment Sequence CABD | Part 3: Treatment Sequence BACE | Part 3: Treatment Sequence ACBE | Part 3: Treatment Sequence CBAE | Part 4: PF-07817883 600 mg (Suspension), Fasted | Part 5: Treatment Sequence AB | Part 5: Treatment Sequence BA | Part 6: Treatment Sequence ABC | Part 6: Treatment Sequence BCA | Part 6: Treatment Sequence CAB | Part 6: Treatment Sequence BAC | Part 6: Treatment Sequence ACB | Part 6: Treatment Sequence CBA
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 (Participants enrolled in Part 5 (sequence AB) of the study.) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 5:SequenceAB:Washout1(Upto 2 Days)
Arm/Group | P1: C1: Placebo,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg, Fast | P1: C1: PF-07817883 150mg,Fast/Placebo,Fast/PF-07817883 4000mg,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/Placebo,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg,Fast | P1: C2: Placebo,Fast/PF-07817883 3000mg,Fast/Placebo,Fed | P1: C2: PF-07817883 500mg,Fast/Placebo,Fast/PF-07817883 500mg,Fed | P1: C2: PF-07817883 500mg,Fast/PF-07817883 3000mg,Fast/PF-07817883 500mg,Fed | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese | Part 3: Treatment Sequence ABCD | Part 3: Treatment Sequence BCAD | Part 3: Treatment Sequence CABD | Part 3: Treatment Sequence BACE | Part 3: Treatment Sequence ACBE | Part 3: Treatment Sequence CBAE | Part 4: PF-07817883 600 mg (Suspension), Fasted | Part 5: Treatment Sequence AB | Part 5: Treatment Sequence BA | Part 6: Treatment Sequence ABC | Part 6: Treatment Sequence BCA | Part 6: Treatment Sequence CAB | Part 6: Treatment Sequence BAC | Part 6: Treatment Sequence ACB | Part 6: Treatment Sequence CBA
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 (Participants who started washout 1 of Part 5 (sequence AB).) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part5:SequenceAB:Period2(up to 10 Days)
Arm/Group | P1: C1: Placebo,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg, Fast | P1: C1: PF-07817883 150mg,Fast/Placebo,Fast/PF-07817883 4000mg,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/Placebo,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg,Fast | P1: C2: Placebo,Fast/PF-07817883 3000mg,Fast/Placebo,Fed | P1: C2: PF-07817883 500mg,Fast/Placebo,Fast/PF-07817883 500mg,Fed | P1: C2: PF-07817883 500mg,Fast/PF-07817883 3000mg,Fast/PF-07817883 500mg,Fed | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese | Part 3: Treatment Sequence ABCD | Part 3: Treatment Sequence BCAD | Part 3: Treatment Sequence CABD | Part 3: Treatment Sequence BACE | Part 3: Treatment Sequence ACBE | Part 3: Treatment Sequence CBAE | Part 4: PF-07817883 600 mg (Suspension), Fasted | Part 5: Treatment Sequence AB | Part 5: Treatment Sequence BA | Part 6: Treatment Sequence ABC | Part 6: Treatment Sequence BCA | Part 6: Treatment Sequence CAB | Part 6: Treatment Sequence BAC | Part 6: Treatment Sequence ACB | Part 6: Treatment Sequence CBA
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 (Participants who started Period 2 of Part 5 (sequence AB).) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part5:Sequence AB:Washout2(up to 7 Days)
Arm/Group | P1: C1: Placebo,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg, Fast | P1: C1: PF-07817883 150mg,Fast/Placebo,Fast/PF-07817883 4000mg,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/Placebo,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg,Fast | P1: C2: Placebo,Fast/PF-07817883 3000mg,Fast/Placebo,Fed | P1: C2: PF-07817883 500mg,Fast/Placebo,Fast/PF-07817883 500mg,Fed | P1: C2: PF-07817883 500mg,Fast/PF-07817883 3000mg,Fast/PF-07817883 500mg,Fed | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese | Part 3: Treatment Sequence ABCD | Part 3: Treatment Sequence BCAD | Part 3: Treatment Sequence CABD | Part 3: Treatment Sequence BACE | Part 3: Treatment Sequence ACBE | Part 3: Treatment Sequence CBAE | Part 4: PF-07817883 600 mg (Suspension), Fasted | Part 5: Treatment Sequence AB | Part 5: Treatment Sequence BA | Part 6: Treatment Sequence ABC | Part 6: Treatment Sequence BCA | Part 6: Treatment Sequence CAB | Part 6: Treatment Sequence BAC | Part 6: Treatment Sequence ACB | Part 6: Treatment Sequence CBA
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 (Participants who started washout 2 of Part 5 (sequence AB).) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part5:Sequence BA:Period1(up to 10 Days)
Arm/Group | P1: C1: Placebo,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg, Fast | P1: C1: PF-07817883 150mg,Fast/Placebo,Fast/PF-07817883 4000mg,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/Placebo,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg,Fast | P1: C2: Placebo,Fast/PF-07817883 3000mg,Fast/Placebo,Fed | P1: C2: PF-07817883 500mg,Fast/Placebo,Fast/PF-07817883 500mg,Fed | P1: C2: PF-07817883 500mg,Fast/PF-07817883 3000mg,Fast/PF-07817883 500mg,Fed | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese | Part 3: Treatment Sequence ABCD | Part 3: Treatment Sequence BCAD | Part 3: Treatment Sequence CABD | Part 3: Treatment Sequence BACE | Part 3: Treatment Sequence ACBE | Part 3: Treatment Sequence CBAE | Part 4: PF-07817883 600 mg (Suspension), Fasted | Part 5: Treatment Sequence AB | Part 5: Treatment Sequence BA | Part 6: Treatment Sequence ABC | Part 6: Treatment Sequence BCA | Part 6: Treatment Sequence CAB | Part 6: Treatment Sequence BAC | Part 6: Treatment Sequence ACB | Part 6: Treatment Sequence CBA
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 (Participants enrolled in Part 5 (sequence BA) of the study.) | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part5:Sequence BA:Washout1(up to 7 Days)
Arm/Group | P1: C1: Placebo,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg, Fast | P1: C1: PF-07817883 150mg,Fast/Placebo,Fast/PF-07817883 4000mg,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/Placebo,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg,Fast | P1: C2: Placebo,Fast/PF-07817883 3000mg,Fast/Placebo,Fed | P1: C2: PF-07817883 500mg,Fast/Placebo,Fast/PF-07817883 500mg,Fed | P1: C2: PF-07817883 500mg,Fast/PF-07817883 3000mg,Fast/PF-07817883 500mg,Fed | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese | Part 3: Treatment Sequence ABCD | Part 3: Treatment Sequence BCAD | Part 3: Treatment Sequence CABD | Part 3: Treatment Sequence BACE | Part 3: Treatment Sequence ACBE | Part 3: Treatment Sequence CBAE | Part 4: PF-07817883 600 mg (Suspension), Fasted | Part 5: Treatment Sequence AB | Part 5: Treatment Sequence BA | Part 6: Treatment Sequence ABC | Part 6: Treatment Sequence BCA | Part 6: Treatment Sequence CAB | Part 6: Treatment Sequence BAC | Part 6: Treatment Sequence ACB | Part 6: Treatment Sequence CBA
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 (Participants who started washout 1 of Part 5 (sequence BA).) | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 5: Sequence BA: Period 2 (Day 1)
Arm/Group | P1: C1: Placebo,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg, Fast | P1: C1: PF-07817883 150mg,Fast/Placebo,Fast/PF-07817883 4000mg,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/Placebo,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg,Fast | P1: C2: Placebo,Fast/PF-07817883 3000mg,Fast/Placebo,Fed | P1: C2: PF-07817883 500mg,Fast/Placebo,Fast/PF-07817883 500mg,Fed | P1: C2: PF-07817883 500mg,Fast/PF-07817883 3000mg,Fast/PF-07817883 500mg,Fed | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese | Part 3: Treatment Sequence ABCD | Part 3: Treatment Sequence BCAD | Part 3: Treatment Sequence CABD | Part 3: Treatment Sequence BACE | Part 3: Treatment Sequence ACBE | Part 3: Treatment Sequence CBAE | Part 4: PF-07817883 600 mg (Suspension), Fasted | Part 5: Treatment Sequence AB | Part 5: Treatment Sequence BA | Part 6: Treatment Sequence ABC | Part 6: Treatment Sequence BCA | Part 6: Treatment Sequence CAB | Part 6: Treatment Sequence BAC | Part 6: Treatment Sequence ACB | Part 6: Treatment Sequence CBA
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 (Participants who started Period 2 of Part 5 (sequence BA).) | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part5:Sequence BA:Washout2(up to 2 Days)
Arm/Group | P1: C1: Placebo,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg, Fast | P1: C1: PF-07817883 150mg,Fast/Placebo,Fast/PF-07817883 4000mg,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/Placebo,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg,Fast | P1: C2: Placebo,Fast/PF-07817883 3000mg,Fast/Placebo,Fed | P1: C2: PF-07817883 500mg,Fast/Placebo,Fast/PF-07817883 500mg,Fed | P1: C2: PF-07817883 500mg,Fast/PF-07817883 3000mg,Fast/PF-07817883 500mg,Fed | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese | Part 3: Treatment Sequence ABCD | Part 3: Treatment Sequence BCAD | Part 3: Treatment Sequence CABD | Part 3: Treatment Sequence BACE | Part 3: Treatment Sequence ACBE | Part 3: Treatment Sequence CBAE | Part 4: PF-07817883 600 mg (Suspension), Fasted | Part 5: Treatment Sequence AB | Part 5: Treatment Sequence BA | Part 6: Treatment Sequence ABC | Part 6: Treatment Sequence BCA | Part 6: Treatment Sequence CAB | Part 6: Treatment Sequence BAC | Part 6: Treatment Sequence ACB | Part 6: Treatment Sequence CBA
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 (Participants who started washout 2 of Part 5 (sequence BA).) | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 6 Period 1 (Day 1)
Arm/Group | P1: C1: Placebo,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg, Fast | P1: C1: PF-07817883 150mg,Fast/Placebo,Fast/PF-07817883 4000mg,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/Placebo,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg,Fast | P1: C2: Placebo,Fast/PF-07817883 3000mg,Fast/Placebo,Fed | P1: C2: PF-07817883 500mg,Fast/Placebo,Fast/PF-07817883 500mg,Fed | P1: C2: PF-07817883 500mg,Fast/PF-07817883 3000mg,Fast/PF-07817883 500mg,Fed | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese | Part 3: Treatment Sequence ABCD | Part 3: Treatment Sequence BCAD | Part 3: Treatment Sequence CABD | Part 3: Treatment Sequence BACE | Part 3: Treatment Sequence ACBE | Part 3: Treatment Sequence CBAE | Part 4: PF-07817883 600 mg (Suspension), Fasted | Part 5: Treatment Sequence AB | Part 5: Treatment Sequence BA | Part 6: Treatment Sequence ABC | Part 6: Treatment Sequence BCA | Part 6: Treatment Sequence CAB | Part 6: Treatment Sequence BAC | Part 6: Treatment Sequence ACB | Part 6: Treatment Sequence CBA
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 (Participants enrolled in Part 6 of the study.) | 4 (Participants enrolled in Part 6 of the study.) | 4 (Participants enrolled in Part 6 of the study.) | 4 (Participants enrolled in Part 6 of the study.) | 4 (Participants enrolled in Part 6 of the study.) | 4 (Participants enrolled in Part 6 of the study.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 6: Washout 1 (up to 7 Days)
Arm/Group | P1: C1: Placebo,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg, Fast | P1: C1: PF-07817883 150mg,Fast/Placebo,Fast/PF-07817883 4000mg,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/Placebo,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg,Fast | P1: C2: Placebo,Fast/PF-07817883 3000mg,Fast/Placebo,Fed | P1: C2: PF-07817883 500mg,Fast/Placebo,Fast/PF-07817883 500mg,Fed | P1: C2: PF-07817883 500mg,Fast/PF-07817883 3000mg,Fast/PF-07817883 500mg,Fed | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese | Part 3: Treatment Sequence ABCD | Part 3: Treatment Sequence BCAD | Part 3: Treatment Sequence CABD | Part 3: Treatment Sequence BACE | Part 3: Treatment Sequence ACBE | Part 3: Treatment Sequence CBAE | Part 4: PF-07817883 600 mg (Suspension), Fasted | Part 5: Treatment Sequence AB | Part 5: Treatment Sequence BA | Part 6: Treatment Sequence ABC | Part 6: Treatment Sequence BCA | Part 6: Treatment Sequence CAB | Part 6: Treatment Sequence BAC | Part 6: Treatment Sequence ACB | Part 6: Treatment Sequence CBA
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 (Participants who started washout 1 of Part 6.) | 4 (Participants who started washout 1 of Part 6.) | 4 (Participants who started washout 1 of Part 6.) | 4 (Participants who started washout 1 of Part 6.) | 4 (Participants who started washout 1 of Part 6.) | 4 (Participants who started washout 1 of Part 6.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 6 Period 2 (Day 1)
Arm/Group | P1: C1: Placebo,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg, Fast | P1: C1: PF-07817883 150mg,Fast/Placebo,Fast/PF-07817883 4000mg,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/Placebo,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg,Fast | P1: C2: Placebo,Fast/PF-07817883 3000mg,Fast/Placebo,Fed | P1: C2: PF-07817883 500mg,Fast/Placebo,Fast/PF-07817883 500mg,Fed | P1: C2: PF-07817883 500mg,Fast/PF-07817883 3000mg,Fast/PF-07817883 500mg,Fed | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese | Part 3: Treatment Sequence ABCD | Part 3: Treatment Sequence BCAD | Part 3: Treatment Sequence CABD | Part 3: Treatment Sequence BACE | Part 3: Treatment Sequence ACBE | Part 3: Treatment Sequence CBAE | Part 4: PF-07817883 600 mg (Suspension), Fasted | Part 5: Treatment Sequence AB | Part 5: Treatment Sequence BA | Part 6: Treatment Sequence ABC | Part 6: Treatment Sequence BCA | Part 6: Treatment Sequence CAB | Part 6: Treatment Sequence BAC | Part 6: Treatment Sequence ACB | Part 6: Treatment Sequence CBA
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 (Participants who started Period 2 of Part 6.) | 4 (Participants who started Period 2 of Part 6.) | 4 (Participants who started Period 2 of Part 6.) | 4 (Participants who started Period 2 of Part 6.) | 4 (Participants who started Period 2 of Part 6.) | 4 (Participants who started Period 2 of Part 6.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 3 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Part 6: Washout 2 (up to 7 Days)
Arm/Group | P1: C1: Placebo,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg, Fast | P1: C1: PF-07817883 150mg,Fast/Placebo,Fast/PF-07817883 4000mg,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/Placebo,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg,Fast | P1: C2: Placebo,Fast/PF-07817883 3000mg,Fast/Placebo,Fed | P1: C2: PF-07817883 500mg,Fast/Placebo,Fast/PF-07817883 500mg,Fed | P1: C2: PF-07817883 500mg,Fast/PF-07817883 3000mg,Fast/PF-07817883 500mg,Fed | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese | Part 3: Treatment Sequence ABCD | Part 3: Treatment Sequence BCAD | Part 3: Treatment Sequence CABD | Part 3: Treatment Sequence BACE | Part 3: Treatment Sequence ACBE | Part 3: Treatment Sequence CBAE | Part 4: PF-07817883 600 mg (Suspension), Fasted | Part 5: Treatment Sequence AB | Part 5: Treatment Sequence BA | Part 6: Treatment Sequence ABC | Part 6: Treatment Sequence BCA | Part 6: Treatment Sequence CAB | Part 6: Treatment Sequence BAC | Part 6: Treatment Sequence ACB | Part 6: Treatment Sequence CBA
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 (Participants who started washout 2 of Part 6.) | 4 (Participants who started washout 2 of Part 6.) | 3 (Participants who started washout 2 of Part 6.) | 4 (Participants who started washout 2 of Part 6.) | 4 (Participants who started washout 2 of Part 6.) | 3 (Participants who started washout 2 of Part 6.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 3 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 6 Period 3 (Day 1)
Arm/Group | P1: C1: Placebo,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg, Fast | P1: C1: PF-07817883 150mg,Fast/Placebo,Fast/PF-07817883 4000mg,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/Placebo,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg,Fast | P1: C2: Placebo,Fast/PF-07817883 3000mg,Fast/Placebo,Fed | P1: C2: PF-07817883 500mg,Fast/Placebo,Fast/PF-07817883 500mg,Fed | P1: C2: PF-07817883 500mg,Fast/PF-07817883 3000mg,Fast/PF-07817883 500mg,Fed | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese | Part 3: Treatment Sequence ABCD | Part 3: Treatment Sequence BCAD | Part 3: Treatment Sequence CABD | Part 3: Treatment Sequence BACE | Part 3: Treatment Sequence ACBE | Part 3: Treatment Sequence CBAE | Part 4: PF-07817883 600 mg (Suspension), Fasted | Part 5: Treatment Sequence AB | Part 5: Treatment Sequence BA | Part 6: Treatment Sequence ABC | Part 6: Treatment Sequence BCA | Part 6: Treatment Sequence CAB | Part 6: Treatment Sequence BAC | Part 6: Treatment Sequence ACB | Part 6: Treatment Sequence CBA
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 (Participants who started Period 3 of Part 6.) | 4 (Participants who started Period 3 of Part 6.) | 3 (Participants who started Period 3 of Part 6.) | 4 (Participants who started Period 3 of Part 6.) | 4 (Participants who started Period 3 of Part 6.) | 3 (Participants who started Period 3 of Part 6.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 3 | 4 | 4 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants were analyzed according to the product they actually received.
Groups:
- Total: Total of all reporting groups
Arm/Group | P1: C1: Placebo,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg, Fast | P1: C1: PF-07817883 150mg,Fast/Placebo,Fast/PF-07817883 4000mg,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/Placebo,Fast | P1: C1: PF-07817883 150 mg,Fast/PF-07817883 1500mg,Fast/PF-07817883 4000mg,Fast | P1: C2: Placebo,Fast/PF-07817883 3000mg,Fast/Placebo,Fed | P1: C2: PF-07817883 500mg,Fast/Placebo,Fast/PF-07817883 500mg,Fed | P1: C2: PF-07817883 500mg,Fast/PF-07817883 3000mg,Fast/PF-07817883 500mg,Fed | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese | Part 3: Treatment Sequence ABCD | Part 3: Treatment Sequence BCAD | Part 3: Treatment Sequence CABD | Part 3: Treatment Sequence BACE | Part 3: Treatment Sequence ACBE | Part 3: Treatment Sequence CBAE | Part 4: PF-07817883 600 mg (Suspension), Fasted | Part 5: Treatment Sequence AB | Part 5: Treatment Sequence BA | Part 6: Treatment Sequence ABC | Part 6: Treatment Sequence BCA | Part 6: Treatment Sequence CAB | Part 6: Treatment Sequence BAC | Part 6: Treatment Sequence ACB | Part 6: Treatment Sequence CBA | Total
Number analyzed (Participants) | 2 | 2 | 2 | 2 | 2 | 2 | 4 | 6 | 4 | 4 | 4 | 1 | 3 | 2 | 2 | 2 | 2 | 2 | 2 | 6 | 7 | 7 | 4 | 4 | 4 | 4 | 4 | 4 | 94
Age, Customized [Count of Participants; unit: Participants] — Data for arm - ''Part 2: Placebo (Suspension) BID, Fasted, Chinese'' is not disclosed to avoid risk of identification and kept under ''Not disclosed'' category.
  Participants
    18-44 Years | 0 | 1 | 1 | 2 | 1 | 1 | 2 | 5 | 2 | 4 | 2 | 0 | 3 | 2 | 0 | 1 | 1 | 2 | 2 | 4 | 4 | 3 | 3 | 4 | 4 | 3 | 3 | 4 | 64
    45-60 Years | 2 | 1 | 1 | 0 | 1 | 1 | 2 | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 2 | 3 | 4 | 1 | 0 | 0 | 1 | 1 | 0 | 29
    Not Disclosed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sex/Gender, Customized [Count of Participants; unit: Participants] — Data for arm - ''Part 2: Placebo (Suspension) BID, Fasted, Chinese'' is not disclosed to avoid risk of identification and kept under ''Not disclosed'' category.
  Participants
    Female | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 2 | 0 | 0 | 2 | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 19
    Male | 1 | 2 | 1 | 2 | 1 | 2 | 3 | 6 | 4 | 2 | 4 | 0 | 3 | 1 | 2 | 0 | 1 | 0 | 2 | 6 | 5 | 5 | 4 | 3 | 3 | 3 | 4 | 4 | 74
    Not Disclosed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Data for arm - ''Part 2: Placebo (Suspension) BID, Fasted, Chinese'' is not disclosed to avoid risk of identification and kept under ''Not disclosed'' category.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
    Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 3 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 4 | 1 | 0 | 1 | 0 | 1 | 1 | 19
    Black or African American | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 3 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 2 | 1 | 1 | 3 | 0 | 1 | 31
    White | 1 | 1 | 1 | 1 | 1 | 1 | 2 | 4 | 1 | 0 | 1 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 1 | 3 | 3 | 2 | 1 | 2 | 2 | 1 | 3 | 2 | 39
    More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
    Not Disclosed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Data for arm - ''Part 2: Placebo (Suspension) BID, Fasted, Chinese'' is not disclosed to avoid risk of identification and kept under ''Not disclosed'' category.
  Participants
    Hispanic or Latino | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 4 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 1 | 3 | 1 | 0 | 3 | 2 | 2 | 2 | 2 | 33
    Not Hispanic or Latino | 1 | 1 | 1 | 1 | 0 | 1 | 3 | 2 | 2 | 4 | 4 | 0 | 3 | 2 | 2 | 0 | 1 | 2 | 2 | 5 | 4 | 6 | 4 | 1 | 2 | 2 | 2 | 2 | 60
    Not Disclosed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE was considered a TEAE if the event started during the effective duration of treatment. All events that started on or after the first dosing day and time/start time, if collected, but before the end of the study were considered as TEAEs.
Time Frame: From start of study treatment up to 28-35 days after administration of last dose of study intervention (maximum up to 48 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Placebo (Suspension), Fasted: Participants who received a single dose of placebo as an oral suspension on Day 1 of either Period 1, 2 or 3 under fasted conditions were included.
- Placebo (Suspension), Fed: Participants who received a single dose of placebo as an oral suspension on Day 1 of either Period 1, 2 or 3 under fed conditions were included.
- PF-07817883 150 mg (Suspension), Fasted: Participants who received a single dose of PF-07817883 150 mg as an oral suspension on Day 1 of either Period 1, 2 or 3 under fasted conditions were included.
- PF-07817883 500 mg (Suspension), Fasted: Participants who received a single dose of PF-07817883 500 mg as an oral suspension on Day 1 of either Period 1, 2 or 3 under fasted conditions were included.
- PF-07817883 500 mg (Suspension), Fed: Participants who received a single dose of PF-07817883 500 mg as an oral suspension on Day 1 of either Period 1, 2 or 3 under fed conditions were included.
- PF-07817883 1500 mg (Suspension), Fasted: Participants who received a single dose of PF-07817883 1500 mg as an oral suspension on Day 1 of either Period 1, 2 or 3 under fasted conditions were included.
- PF-07817883 3000 mg (Suspension), Fasted: Participants who received a single dose of PF-07817883 3000 mg as an oral suspension on Day 1 of either Period 1, 2 or 3 under fasted conditions were included.
- PF-07817883 4000 mg (Suspension), Fasted: Participants who received a single dose of PF-07817883 4000 mg as an oral suspension on Day 1 of either Period 1, 2 or 3 under fasted conditions were included.
Arm/Group | Placebo (Suspension), Fasted | Placebo (Suspension), Fed | PF-07817883 150 mg (Suspension), Fasted | PF-07817883 500 mg (Suspension), Fasted | PF-07817883 500 mg (Suspension), Fed | PF-07817883 1500 mg (Suspension), Fasted | PF-07817883 3000 mg (Suspension), Fasted | PF-07817883 4000 mg (Suspension), Fasted
Number analyzed (Participants) | 10 | 2 | 6 | 6 | 4 | 6 | 5 | 5
Participants | 4 | 1 | 2 | 1 | 0 | 3 | 0 | 1

2. Primary Outcome: Part 1: Number of Participants With Laboratory Test Abnormalities
Description: Laboratory parameters included: (lymphocytes less than (<) 0.8*lower limit of normal [LLN] [10^3 per millimeter cube {mm3}], lymphocytes/leukocytes <0.8*LLN [percentage {%}], neutrophils <0.8*LLN [10^3/mm3], neutrophils/leukocytes <0.8*LLN [%], monocytes/leukocytes greater than (>) 1.2*upper limit of normal [ULN] [%], partial thromboplastin time >1.1*ULN [seconds]), chemistry (bicarbonate <0.9*LLN [milliequivalents per liter {mEq/L}], creatine kinase >2.0*ULN [units per liter {U/L}], lipase >1.5*ULN [U/L]), and urinalysis (urine hemoglobin greater than or equal to [>=] 1, leukocyte esterase >=1). Number of participants with any lab test abnormalities meeting the pre-specified criteria are reported in this outcome measure.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Suspension), Fasted | Placebo (Suspension), Fed | PF-07817883 150 mg (Suspension), Fasted | PF-07817883 500 mg (Suspension), Fasted | PF-07817883 500 mg (Suspension), Fed | PF-07817883 1500 mg (Suspension), Fasted | PF-07817883 3000 mg (Suspension), Fasted | PF-07817883 4000 mg (Suspension), Fasted
Number analyzed (Participants) | 10 | 2 | 6 | 6 | 4 | 6 | 5 | 5
Participants | 5 | 1 | 2 | 2 | 1 | 1 | 2 | 2

3. Primary Outcome: Part 1: Number of Participants With Vital Signs Meeting Pre-Defined Criteria
Description: Vital signs including systolic blood pressure (SBP), diastolic blood pressure (DBP) and pulse rate (PR) were measured in a supine position after approximately 5 minutes of rest for the participant. Criteria for vital signs included: SBP: value less than (<) 90 millimeter of mercury (mmHg), change greater than or equal to (>=) 30 mmHg increase, change >= 30 mmHg decrease; DBP: value < 50 mmHg, change >= 20 mmHg increase, change >= 20 mmHg decrease; PR: value < 40 beats per minute (bpm), value > 120 bpm.
Time Frame: Up to Day 2 of each period
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Suspension), Fasted | Placebo (Suspension), Fed | PF-07817883 150 mg (Suspension), Fasted | PF-07817883 500 mg (Suspension), Fasted | PF-07817883 500 mg (Suspension), Fed | PF-07817883 1500 mg (Suspension), Fasted | PF-07817883 3000 mg (Suspension), Fasted | PF-07817883 4000 mg (Suspension), Fasted
Number analyzed (Participants) | 10 | 2 | 6 | 6 | 4 | 6 | 5 | 5
Participants
  SBP value < 90 mmHg | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
  SBP Change >= 30 mmHg increase | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  SBP Change >= 30 mmHg decrease | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
  DBP Value < 50 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DBP Change >= 20 mmHg increase | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  DBP Change >= 20 mmHg decrease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR Value < 40 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR Value > 120 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Part 1: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: Standard 12 lead ECGs were obtained with the participant in a supine position after at least 5 minutes of rest using an ECG machine that automatically calculated the heart rate and measured PR interval, QT interval, QTcF and QRS complex. Number of participants with abnormalities in ECG were reported in this outcome measure.
Time Frame: Up to Day 2 of each period
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Suspension), Fasted | Placebo (Suspension), Fed | PF-07817883 150 mg (Suspension), Fasted | PF-07817883 500 mg (Suspension), Fasted | PF-07817883 500 mg (Suspension), Fed | PF-07817883 1500 mg (Suspension), Fasted | PF-07817883 3000 mg (Suspension), Fasted | PF-07817883 4000 mg (Suspension), Fasted
Number analyzed (Participants) | 10 | 2 | 6 | 6 | 4 | 6 | 5 | 5
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Primary Outcome: Part 2: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a participant temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE was considered a TEAE if the event started during the effective duration of treatment. All events that started on or after the first dosing day and time/start time, if collected, but before the end of the study were considered as TEAEs.
Time Frame: From start of study treatment up to 38-45 days after administration of last dose of study intervention (maximum up to 55 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese
Number analyzed (Participants) | 6 | 4 | 4 | 4 | 1 | 3
Participants | 2 | 1 | 0 | 2 | 0 | 2

6. Primary Outcome: Part 2: Number of Participants With Laboratory Test Abnormalities
Description: Laboratory parameters included: hematology (lymphocytes/leukocytes >1.2*ULN [%], neutrophils <0.8*LLN [10^3/mm3], neutrophils/leukocytes <0.8*LLN [%], monocytes/leukocytes >1.2*ULN [%]), chemistry (urate >1.2*ULN [milligrams per deciliter] {mg/dL}), and urinalysis (ketones >=1, urine hemoglobin >=1). Number of participants with any lab test abnormalities meeting the pre-specified criteria are reported in this outcome measure.
Time Frame: as for outcome 5
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese
Number analyzed (Participants) | 6 | 4 | 4 | 4 | 1 | 3
Participants | 1 | 2 | 2 | 2 | 0 | 1

7. Primary Outcome: Part 2: Number of Participants With Vital Signs Meeting Pre-Defined Criteria
Description: Vital signs including SBP, DBP and PR were measured in a supine position after approximately 5 minutes of rest for the participant. Criteria for vital signs included: SBP: value < 90 mmHg, change >= 30 mmHg increase, change >= 30 mmHg decrease; DBP: value < 50 mmHg, change >= 20 mmHg increase, change >= 20 mmHg decrease; PR: value < 40 bpm, value > 120 bpm. 4. Number of participants with vital signs meeting any of the pre-defined criteria is reported in this outcome measure.
Time Frame: Up to Day 12
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese
Number analyzed (Participants) | 6 | 4 | 4 | 4 | 1 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Part 2: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: as for outcome 4
Time Frame: Up to Day 12
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese
Number analyzed (Participants) | 6 | 4 | 4 | 4 | 1 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0

9. Primary Outcome: Part 3:Ratio Based on Area Under Plasma Concentration Time Curve From Time 0 to Time of Last Quantifiable Concentration (AUClast) and Area Under Concentration-Time Curve From Time 0 Extrapolated to Infinite Time (AUCinf) of Oral Formulation and Suspension
Description: Data for AUClast and AUCinf are reported in the descriptive section. AUClast was calculated by the linear/log trapezoidal method. AUCinf was calculated as AUClast + (Clast/kel), where Clast was the predicted plasma concentration at the last quantifiable time point from the log-linear regression analysis. Ratio based on AUClast and AUCinf of oral formulation and suspension were reported in statistical analysis.
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 hours post-dose)
Population: Pharmacokinetic (PK) parameter set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of interest were reported. Here, ''Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*Hour per milliliter (ng*hr/mL)
Groups:
- Part 3: PF-07817883 600 mg (Suspension), Fasted: Participants received a single dose of PF-07817883 600 mg oral suspension under fasted conditions on Day 1 of either Period 1, 2, 3 or 4. An overnight fast for approximately 10 hours was required.
- Part 3: PF-07817883 SDD 600 mg (Tablet), Fasted: Participants received a single dose of PF-07817883 600 mg spray dried dispersion (SDD) under fasted conditions on Day 1 of either Period 1, 2, 3 or 4. An overnight fast for approximately 10 hours was required.
- Part 3: PF-07817883 SDD 600 mg (Tablet), Fed: Participants received a single dose of PF-07817883 600 mg spray dried dispersion (SDD) under fed conditions on Day 1 of either Period 1, 2, 3 or 4. PF-07817883 was administered approximately 10 minutes after finishing the meal/snack.
- Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fasted: Participants received a single dose of PF-07817883 600 mg crystalline tablet under fasted conditions on Day 1 of either Period 1, 2, 3 or 4. An overnight fast for approximately 10 hours was required.
- Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fed: Participants received a single dose of PF-07817883 600 mg crystalline tablet under fed conditions on Day 1 of either Period 1, 2, 3 or 4. PF-07817883 was administered approximately 10 minutes after finishing the meal/snack.
Arm/Group | Part 3: PF-07817883 600 mg (Suspension), Fasted | Part 3: PF-07817883 SDD 600 mg (Tablet), Fasted | Part 3: PF-07817883 SDD 600 mg (Tablet), Fed | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fasted | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fed
Number analyzed (Participants) | 12 | 12 | 6 | 12 | 6
Nanogram*Hour per milliliter (ng*hr/mL)
  AUCinf: number analyzed (Participants) | 12 | 12 | 6 | 11 | 4
  AUCinf | 42970 (35) | 44140 (38) | 28430 (28) | 42930 (43) | 46170 (27)
  AUClast | 42540 (35) | 43570 (37) | 27750 (29) | 41620 (41) | 35930 (54)
Statistical Analysis 1: Comparison: Part 3: PF-07817883 600 mg (Suspension), Fasted vs Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fasted; AUCinf; Test type: Other; Ratio of Adjusted Geometric Means = 101.29, 90% CI 2-sided [95.71 to 107.18] — A mixed effect model was used with sequence, period and treatment as fixed effect and participant nested within sequence as random effect. Values had been back-transformed from natural log scale. Ratios (and 90% CIs) were expressed as percentages
Statistical Analysis 2: Comparison: Part 3: PF-07817883 600 mg (Suspension), Fasted vs Part 3: PF-07817883 SDD 600 mg (Tablet), Fasted; AUCinf; Test type: Other; Ratio of Adjusted Geometric Means = 102.74, 90% CI 2-sided [97.28 to 108.50] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Part 3: PF-07817883 600 mg (Suspension), Fasted vs Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fasted; AUClast; Test type: Other; Ratio of Adjusted Geometric Means = 97.83, 90% CI 2-sided [91.32 to 104.80] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 4: Comparison: Part 3: PF-07817883 600 mg (Suspension), Fasted vs Part 3: PF-07817883 SDD 600 mg (Tablet), Fasted; AUClast; Test type: Other; Ratio of Adjusted Geometric Means = 102.41, 90% CI 2-sided [95.60 to 109.70] — [estimate comment as in outcome 9, analysis 1]

10. Primary Outcome: Part 3: Ratio Based on Maximum Observed Concentration (Cmax) of Oral Formulation and Suspension
Description: Data for Cmax are reported in the descriptive section. Ratio based on Cmax of oral formulation and suspension were reported in statistical analysis.
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 hours post-dose)
Population: PK parameter set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of interest were reported.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Part 3: PF-07817883 600 mg (Suspension), Fasted | Part 3: PF-07817883 SDD 600 mg (Tablet), Fasted | Part 3: PF-07817883 SDD 600 mg (Tablet), Fed | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fasted | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fed
Number analyzed (Participants) | 12 | 12 | 6 | 12 | 6
Nanogram per milliliter (ng/mL) | 9354 (18) | 6934 (35) | 4590 (21) | 6284 (38) | 5008 (47)
Statistical Analysis 1: Comparison: Part 3: PF-07817883 600 mg (Suspension), Fasted vs Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fasted; Test type: Other; Ratio of Adjusted Geometric Means = 67.18, 90% CI 2-sided [58.13 to 77.65] — [estimate comment as in outcome 9, analysis 1]
Statistical Analysis 2: Comparison: Part 3: PF-07817883 600 mg (Suspension), Fasted vs Part 3: PF-07817883 SDD 600 mg (Tablet), Fasted; Test type: Other; Ratio of Adjusted Geometric Means = 74.12, 90% CI 2-sided [64.14 to 85.67] — [estimate comment as in outcome 9, analysis 1]

11. Primary Outcome: Part 4: Percentage of Total Dose Administered Recovered in Urine
Description: The percentage of total dose administered recovered in urine was reported in this outcome measure.
Time Frame: Up to 144 hours post-dose
Population: PK parameter set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of interest were reported. Here, ''Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percentage dose excreted
Arm/Group | Part 4: PF-07817883 600 mg (Suspension), Fasted
Number analyzed (Participants) | 4
Percentage dose excreted | 12.6 (4.7)

12. Primary Outcome: Part 4: Percentage of Total Dose Administered Recovered in Feces
Description: The percentage of total dose administered recovered in feces was reported in this outcome measure.
Time Frame: Up to 144 hours post-dose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percentage dose excreted
Arm/Group | Part 4: PF-07817883 600 mg (Suspension), Fasted
Number analyzed (Participants) | 4
Percentage dose excreted | 88.9 (10)

13. Primary Outcome: Part 4: Percentage of Total Dose Administered Recovered in Urine and Feces
Description: The percentage of total dose administered recovered in urine and feces was reported in this outcome measure.
Time Frame: Up to 144 hours post-dose
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Percentage dose excreted
Arm/Group | Part 4: PF-07817883 600 mg (Suspension), Fasted
Number analyzed (Participants) | 4
Percentage dose excreted | 101.5 (7.7)

14. Primary Outcome: Part 5: Maximum Observed Concentration (Cmax) of Midazolam
Description: Cmax of midazolam was reported in this outcome measure.
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose) for Midazolam 5 mg arm and Day 10 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 36, 48 hours post-dose) for PF-07817883 600 mg (Suspension) BID/ Midazolam 5 mg arm
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Groups:
- PF-07817883 600 mg (Suspension) BID/ Midazolam 5 mg: Participants received PF-07817883 600 mg oral suspension twice a day (BID) for 10 days (Day 1 morning to Day 10 morning). On Day 10 morning, participants received a single oral dose of 5 mg midazolam administered with PF-07817883.
- Midazolam 5 mg: Participants received oral solution of Midazolam 5 mg on Day 1 of either Period 1 or 2.
Arm/Group | PF-07817883 600 mg (Suspension) BID/ Midazolam 5 mg | Midazolam 5 mg
Number analyzed (Participants) | 12 | 13
Nanogram per milliliter (ng/mL) | 33.71 (34) | 30.20 (28)

15. Primary Outcome: Part 5: Area Under the Concentration -Time Curve From Time Zero (0) Extrapolated to Infinite Time (AUCinf) of Midazolam
Description: AUCinf of midazolam was reported in this outcome measure. AUCinf was calculated as AUClast + (Clast/kel), where Clast was the predicted plasma concentration at the last quantifiable time point from the log-linear regression analysis.
Time Frame: as for outcome 14
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*Hour per milliliter (ng*hr/mL)
Arm/Group | PF-07817883 600 mg (Suspension) BID/ Midazolam 5 mg | Midazolam 5 mg
Number analyzed (Participants) | 12 | 13
Nanogram*Hour per milliliter (ng*hr/mL) | 94.30 (26) | 79.85 (31)

16. Primary Outcome: Part 6: Number of Participants With TEAEs
Description: as for outcome 5
Time Frame: From start of study treatment up to 28-35 days after administration of last dose of study intervention (maximum up to 52 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Placebo (Suspension), Fasted: Participants received Placebo oral suspension at 0 and 1 hours on Day 1 of either Period 1, 2 or 3 following an overnight fast of at least 10 hours.
- PF-07817883 6000 mg (Suspension), Fasted: Participants received 6000 mg PF-07817883 oral suspension administered as two split doses of 3000 mg at 0 and 1 hour on Day 1 of either Period 1, 2 or 3 following an overnight fast of at least 10 hours.
- Moxifloxacin 400 mg, Fasted: Participants received 400 mg Moxifloxacin oral tablet and placebo at 0 and 1 hour respectively on Day 1 of either Period 1, 2 or 3 following an overnight fast of at least 10 hours.
Arm/Group | Placebo (Suspension), Fasted | PF-07817883 6000 mg (Suspension), Fasted | Moxifloxacin 400 mg, Fasted
Number analyzed (Participants) | 23 | 23 | 24
Participants | 4 | 6 | 4

17. Primary Outcome: Part 6: Number of Participants With Laboratory Test Abnormalities
Description: Laboratory parameters included: hematology (lymphocytes <0.6*LLN [10^3/mm3], lymphocytes/leukocytes >1.2*ULN [%], neutrophils <0.8*LLN [10^3/mm3], neutrophils/leukocytes <0.8*LLN [%], basophils/leukocytes >1.2*ULN [%], eosinophils/leukocytes >1.2*ULN [%], monocytes/leukocytes >1.2*ULN [%], partial thromboplastin time >1.1*ULN [seconds], prothrombin time >1.1*ULN [seconds]), chemistry (bicarbonate <0.9*LLN [mEq/L], creatine kinase > 2.0*ULN [U/L], lipase > 1.5*ULN [U/L], urobilinogen >=1 [ehrlich units/deciliter] {EU/dL}) and urinalysis (urine hemoglobin >=1, leukocyte esterase >=1, ketones >=1, bacteria >20 [per low power field] {/lpf}). Number of participants with any lab test abnormalities meeting the pre-specified criteria are reported in this outcome measure.
Time Frame: as for outcome 16
Population: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants were analyzed according to the product they actually received. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Suspension), Fasted | PF-07817883 6000 mg (Suspension), Fasted | Moxifloxacin 400 mg, Fasted
Number analyzed (Participants) | 23 | 22 | 24
Participants | 12 | 12 | 7

18. Primary Outcome: Part 6: Number of Participants With Vital Signs Meeting Pre-Defined Criteria
Description: Vital signs including SBP, DBP and PR were measured in a supine position after approximately 5 minutes of rest for the participant. Criteria for vital signs included: SBP: value < 90 mmHg, change >= 30 mmHg increase, change >= 30 mmHg decrease; DBP: value < 50 mmHg, change >= 20 mmHg increase, change >= 20 mmHg decrease; PR: value < 40 bpm, value > 120 bpm.
Time Frame: Up to Day 6 of each period
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Suspension), Fasted | PF-07817883 6000 mg (Suspension), Fasted | Moxifloxacin 400 mg, Fasted
Number analyzed (Participants) | 23 | 23 | 24
Participants
  SBP value < 90 mmHg | 1 | 2 | 3
  SBP change >= 30 mmHg increase | 0 | 1 | 0
  SBP change >= 30 mmHg decrease | 0 | 0 | 0
  DBP value < 50 mmHg | 0 | 0 | 0
  DBP change >= 20 mmHg increase | 0 | 0 | 0
  DBP change >= 20 mmHg decrease | 0 | 0 | 1
  Pulse rate value < 40 bpm | 0 | 0 | 0
  Pulse rate value > 120 bpm | 0 | 0 | 0

19. Primary Outcome: Part 6: Number of Participants According to Categorization of ECG Data
Description: Standard 12 lead ECGs were obtained with the participant in a supine position after at least 5 minutes of rest using an ECG machine that automatically calculated the heart rate and measured QTcF interval, aggregate 450 milliseconds (msec) < value <= 480 msec and QTcF interval, aggregate 30 msec < change <= 60 msec. Number of participants with abnormalities in ECG were reported in this outcome measure.
Time Frame: Up to Day 6 of each period
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Suspension), Fasted | PF-07817883 6000 mg (Suspension), Fasted | Moxifloxacin 400 mg, Fasted
Number analyzed (Participants) | 23 | 23 | 24
Participants
  QTCF interval, aggregate 450 msec < Value <= 480 msec | 0 | 0 | 1
  QTCF interval, aggregate 30 msec < Change <= 60 msec | 0 | 0 | 1

20. Secondary Outcome: Part 1: Maximum Observed Concentration (Cmax) of PF-07817883
Description: Cmax of PF-07817883 was reported in this outcome measure.
Time Frame: Day 1 (pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48, 72 hours post-dose)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | PF-07817883 150 mg (Suspension), Fasted | PF-07817883 500 mg (Suspension), Fasted | PF-07817883 500 mg (Suspension), Fed | PF-07817883 1500 mg (Suspension), Fasted | PF-07817883 3000 mg (Suspension), Fasted | PF-07817883 4000 mg (Suspension), Fasted
Number analyzed (Participants) | 6 | 6 | 4 | 6 | 5 | 5
Nanogram per milliliter (ng/mL) | 2269 (51) | 6235 (20) | 3223 (13) | 17420 (36) | 34420 (12) | 34670 (36)

21. Secondary Outcome: Part 1: Time for Cmax (Tmax) of PF-07817883
Description: Tmax of PF-07817883 was reported in this outcome measure.
Time Frame: Day 1 (pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48, 72 hours post-dose)
Population: as for outcome 10
Measure: Median (Full Range); unit: Hours
Arm/Group | PF-07817883 150 mg (Suspension), Fasted | PF-07817883 500 mg (Suspension), Fasted | PF-07817883 500 mg (Suspension), Fed | PF-07817883 1500 mg (Suspension), Fasted | PF-07817883 3000 mg (Suspension), Fasted | PF-07817883 4000 mg (Suspension), Fasted
Number analyzed (Participants) | 6 | 6 | 4 | 6 | 5 | 5
Hours | 1.00 [0.500 to 1.50] | 0.792 [0.500 to 1.50] | 1.25 [1.00 to 2.00] | 0.500 [0.500 to 1.00] | 0.500 [0.500 to 1.05] | 1.00 [0.550 to 1.50]

22. Secondary Outcome: Part 1: Area Under Plasma Concentration Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of PF-07817883
Description: AUClast of PF-07817883 was reported in this outcome measure. AUClast was calculated by the linear/log trapezoidal method.
Time Frame: Day 1 (pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48, 72 hours post-dose)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter
Arm/Group | PF-07817883 150 mg (Suspension), Fasted | PF-07817883 500 mg (Suspension), Fasted | PF-07817883 500 mg (Suspension), Fed | PF-07817883 1500 mg (Suspension), Fasted | PF-07817883 3000 mg (Suspension), Fasted | PF-07817883 4000 mg (Suspension), Fasted
Number analyzed (Participants) | 6 | 6 | 4 | 6 | 5 | 5
Nanogram*hour per milliliter | 10890 (47) | 34580 (25) | 27080 (25) | 83490 (36) | 160700 (33) | 185700 (17)

23. Secondary Outcome: Part 1: Dose Normalized Cmax (Cmax[dn]) of PF-07817883
Description: Cmax(dn) of PF-07817883 was reported in this outcome measure. Cmax(dn) was calculated as Cmax/dose.
Time Frame: Day 1 (pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48, 72 hours post-dose)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter per milligram
Arm/Group | PF-07817883 150 mg (Suspension), Fasted | PF-07817883 500 mg (Suspension), Fasted | PF-07817883 500 mg (Suspension), Fed | PF-07817883 1500 mg (Suspension), Fasted | PF-07817883 3000 mg (Suspension), Fasted | PF-07817883 4000 mg (Suspension), Fasted
Number analyzed (Participants) | 6 | 6 | 4 | 6 | 5 | 5
Nanogram per milliliter per milligram | 15.14 (51) | 12.48 (19) | 6.445 (13) | 11.61 (36) | 11.49 (12) | 8.672 (36)

24. Secondary Outcome: Part 1: Dose Normalized AUClast (AUClast[dn]) of PF-07817883
Description: AUClast(dn) of PF-07817883 was reported in this outcome measure. AUClast(dn) was calculated by AUClast/dose.
Time Frame: Day 1 (pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48, 72 hours post-dose)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour/milliliter/milligram
Arm/Group | PF-07817883 150 mg (Suspension), Fasted | PF-07817883 500 mg (Suspension), Fasted | PF-07817883 500 mg (Suspension), Fed | PF-07817883 1500 mg (Suspension), Fasted | PF-07817883 3000 mg (Suspension), Fasted | PF-07817883 4000 mg (Suspension), Fasted
Number analyzed (Participants) | 6 | 6 | 4 | 6 | 5 | 5
Nanogram*hour/milliliter/milligram | 72.61 (47) | 69.17 (25) | 54.16 (25) | 55.64 (35) | 53.53 (33) | 46.43 (17)

25. Secondary Outcome: Part 1: Area Under the Concentration -Time Curve From Time Zero (0) Extrapolated to Infinite Time (AUCinf) of PF-07817883
Description: AUCinf of PF-07817883 was reported in this outcome measure. AUCinf was calculated as AUClast + (Clast/kel), where Clast was the predicted plasma concentration at the last quantifiable time point from the log-linear regression analysis.
Time Frame: Day 1 (pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48, 72 hours post-dose)
Population: PK parameter set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of interest were reported. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | PF-07817883 150 mg (Suspension), Fasted | PF-07817883 500 mg (Suspension), Fasted | PF-07817883 500 mg (Suspension), Fed | PF-07817883 1500 mg (Suspension), Fasted | PF-07817883 3000 mg (Suspension), Fasted | PF-07817883 4000 mg (Suspension), Fasted
Number analyzed (Participants) | 5 | 6 | 4 | 6 | 5 | 5
Nanogram*hour/milliliter (ng*hr/mL) | 11250 (53) | 35950 (25) | 28120 (28) | 85320 (34) | 166100 (34) | 189400 (19)

26. Secondary Outcome: Part 1: Dose Normalized AUCinf (AUCinf[dn]) of PF-07817883
Description: AUCinf(dn) of PF-07817883 was reported in this outcome measure. AUCinf(dn) was calculated as AUCinf/dose.
Time Frame: Day 1 (pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48, 72 hours post-dose)
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour/milliliter/milligram
Arm/Group | PF-07817883 150 mg (Suspension), Fasted | PF-07817883 500 mg (Suspension), Fasted | PF-07817883 500 mg (Suspension), Fed | PF-07817883 1500 mg (Suspension), Fasted | PF-07817883 3000 mg (Suspension), Fasted | PF-07817883 4000 mg (Suspension), Fasted
Number analyzed (Participants) | 5 | 6 | 4 | 6 | 5 | 5
Nanogram*hour/milliliter/milligram | 74.99 (53) | 71.81 (25) | 56.23 (28) | 56.86 (34) | 55.33 (35) | 47.34 (19)

27. Secondary Outcome: Part 1: Terminal Half-Life (t1/2) of PF-07817883
Description: t1/2 of PF-07817883 was reported in this outcome measure. t1/2 was calculated by Loge(2)/kel, where kel was the terminal phase rate constant calculated by a linear regression of the log linear concentration-time curve. Only those data points judged to describe the terminal log-linear decline were used in the regression.
Time Frame: Day 1 (pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48, 72 hours post-dose)
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | PF-07817883 150 mg (Suspension), Fasted | PF-07817883 500 mg (Suspension), Fasted | PF-07817883 500 mg (Suspension), Fed | PF-07817883 1500 mg (Suspension), Fasted | PF-07817883 3000 mg (Suspension), Fasted | PF-07817883 4000 mg (Suspension), Fasted
Number analyzed (Participants) | 5 | 6 | 4 | 6 | 5 | 5
Hours | 4.534 (0.50659) | 13.88 (10.838) | 15.95 (8.4657) | 10.84 (6.1747) | 18.79 (14.234) | 13.05 (7.3974)

28. Secondary Outcome: Part 1: Apparent Volume of Distribution (Vz/F) of PF-07817883
Description: Vz/F of PF-07817883 was reported in this outcome measure. Vz/F was calculated as dose/(AUCinf*kel).
Time Frame: Day 1 (pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48, 72 hours post-dose)
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter (L)
Arm/Group | PF-07817883 150 mg (Suspension), Fasted | PF-07817883 500 mg (Suspension), Fasted | PF-07817883 500 mg (Suspension), Fed | PF-07817883 1500 mg (Suspension), Fasted | PF-07817883 3000 mg (Suspension), Fasted | PF-07817883 4000 mg (Suspension), Fasted
Number analyzed (Participants) | 5 | 6 | 4 | 6 | 5 | 5
Liter (L) | 86.87 (48) | 209.5 (101) | 366.1 (50) | 242.9 (80) | 367.4 (87) | 358.7 (44)

29. Secondary Outcome: Part 1: Apparent Clearance (CL/F) of PF-07817883
Description: CL/F of PF-07817883 was reported in this outcome measure. CL/F was calculated as dose/AUCinf.
Time Frame: Day 1 (pre-dose, 0.25, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48, 72 hours post-dose)
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter per hour (L/hr)
Arm/Group | PF-07817883 150 mg (Suspension), Fasted | PF-07817883 500 mg (Suspension), Fasted | PF-07817883 500 mg (Suspension), Fed | PF-07817883 1500 mg (Suspension), Fasted | PF-07817883 3000 mg (Suspension), Fasted | PF-07817883 4000 mg (Suspension), Fasted
Number analyzed (Participants) | 5 | 6 | 4 | 6 | 5 | 5
Liter per hour (L/hr) | 13.33 (53) | 13.93 (25) | 17.79 (28) | 17.58 (35) | 18.09 (35) | 21.13 (19)

30. Secondary Outcome: Part 2: Maximum Observed Concentration (Cmax) of PF-07817883 on Days 1, 5 and 10
Description: Cmax of PF-07817883 was reported in this outcome measure.
Time Frame: Day 1 and Day 5 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12 hours post-dose) and Day 10 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 hours post-dose)
Population: PK parameter set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of interest were reported. Here, ''Number Analyzed'' signifies participants evaluable at specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter
Arm/Group | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese
Number analyzed (Participants) | 4 | 4 | 4 | 3
Nanogram/milliliter
  Day 1 | 3582 (20) | 8470 (39) | 24100 (22) | 8381 (12)
  Day 5 | 4234 (7) | 9112 (14) | 27530 (22) | 8260 (18)
  Day 10: number analyzed (Participants) | 4 | 3 | 4 | 3
  Day 10 | 3492 (15) | 7852 (21) | 23420 (14) | 7306 (25)

31. Secondary Outcome: Part 2: Time for Cmax (Tmax) of PF-07817883 on Days 1, 5 and 10
Description: Tmax of PF-07817883 was reported in this outcome measure.
Time Frame: as for outcome 30
Population: as for outcome 30
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese
Number analyzed (Participants) | 4 | 4 | 4 | 3
Hours
  Day 1 | 0.759 [0.500 to 1.00] | 0.775 [0.500 to 1.00] | 0.500 [0.500 to 1.50] | 1.00 [1.00 to 1.05]
  Day 5 | 0.859 [0.500 to 1.02] | 0.500 [0.500 to 0.500] | 0.500 [0.500 to 1.00] | 0.500 [0.500 to 1.00]
  Day 10: number analyzed (Participants) | 4 | 3 | 4 | 3
  Day 10 | 0.500 [0.500 to 1.00] | 0.500 [0.500 to 1.00] | 0.500 [0.500 to 0.500] | 0.533 [0.500 to 1.00]

32. Secondary Outcome: Part 2: Area Under the Plasma Concentration-Time Profile From Time 0 to Time Tau, the Dosing Interval (AUCtau) of PF-07817883 on Days 1, 5 and 10
Description: AUCtau was defined as area under the plasma concentration-time profile from time 0 to time tau, the dosing interval, where tau= 12 hours. AUCtau of PF-07817883 was reported in this outcome measure. AUCtau was calculated by linear/log trapezoidal method.
Time Frame: Day 1 and Day 5 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12 hours post-dose) and Day 10 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12 hours post-dose)
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese
Number analyzed (Participants) | 4 | 4 | 4 | 3
Nanogram*hour per milliliter (ng*hr/mL)
  Day 1 | 14760 (26) | 36440 (27) | 108400 (15) | 36880 (22)
  Day 5 | 18460 (15) | 36300 (10) | 114000 (22) | 37680 (29)
  Day 10: number analyzed (Participants) | 4 | 3 | 4 | 3
  Day 10 | 17180 (10) | 34960 (8) | 103900 (18) | 34650 (29)

33. Secondary Outcome: Part 2: Concentration at 12 Hour Nominal Time Post-Dose (C12) of PF-07817883 on Days 5 and 10
Description: C12 of PF-07817883 was reported in this outcome measure.
Time Frame: 12 hours on Day 5 and Day 10
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese
Number analyzed (Participants) | 4 | 4 | 4 | 3
Nanogram per milliliter (ng/mL)
  Day 5 | 389.3 (15) | 734.5 (15) | 2598 (47) | 716.0 (47)
  Day 10: number analyzed (Participants) | 4 | 3 | 4 | 3
  Day 10 | 425.7 (12) | 865.9 (22) | 2315 (35) | 585.5 (28)

34. Secondary Outcome: Part 2: Dose Normalized Cmax (Cmax[dn]) of PF-07817883 on Days 1, 5 and 10
Description: Cmax(dn) of PF-07817883 was reported in this outcome measure. Cmax(dn) was calculated as Cmax/dose.
Time Frame: as for outcome 30
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter/milligram (ng/mL/mg)
Arm/Group | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese
Number analyzed (Participants) | 4 | 4 | 4 | 3
Nanogram/milliliter/milligram (ng/mL/mg)
  Day 1 | 17.93 (20) | 14.15 (39) | 16.07 (22) | 14.00 (12)
  Day 5 | 21.18 (7) | 15.20 (13) | 18.35 (22) | 13.76 (18)
  Day 10: number analyzed (Participants) | 4 | 3 | 4 | 3
  Day 10 | 17.47 (15) | 13.07 (21) | 15.61 (14) | 12.20 (25)

35. Secondary Outcome: Part 2: Dose Normalized AUCtau (AUCtau[dn]) of PF-07817883 on Days 1, 5 and 10
Description: AUCtau(dn) was defined as dose normalized AUCtau, where tau= 12 hours. AUCtau(dn) of PF-07817883 was reported in this outcome measure. AUCtau(dn) was calculated as AUCtau/dose.
Time Frame: as for outcome 32
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour/milliliter/milligram
Arm/Group | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese
Number analyzed (Participants) | 4 | 4 | 4 | 3
Nanogram*hour/milliliter/milligram
  Day 1 | 73.94 (26) | 60.70 (27) | 72.25 (15) | 61.44 (22)
  Day 5 | 92.46 (15) | 60.49 (10) | 76.20 (23) | 62.82 (29)
  Day 10: number analyzed (Participants) | 4 | 3 | 4 | 3
  Day 10 | 86.04 (10) | 58.28 (8) | 69.43 (18) | 57.78 (29)

36. Secondary Outcome: Part 2: Average Concentration (Cav) of PF-07817883 on Days 5 and 10
Description: Cav of PF-07817883 was reported in this outcome measure. Cav was calculated as AUCtau/12.
Time Frame: Day 5 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12 hours post-dose) and Day 10 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12 hours post-dose)
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter (ng/mL)
Arm/Group | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese
Number analyzed (Participants) | 4 | 4 | 4 | 3
Nanogram/milliliter (ng/mL)
  Day 5 | 1542 (15) | 3022 (10) | 9515 (22) | 3140 (29)
  Day 10: number analyzed (Participants) | 4 | 3 | 4 | 3
  Day 10 | 1434 (10) | 2914 (8) | 8672 (18) | 2890 (29)

37. Secondary Outcome: Part 2: Observed Accumulation Ratio for AUCtau (Rac) of PF-07817883 on Days 5 and 10
Description: Rac was defined as observed accumulation ratio for AUCtau, where tau= 12 hours. Rac of PF-07817883 was reported in this outcome measure. Rac was calculated as AUCtau on Day 5 or Day 10/AUCtau on Day 1.
Time Frame: as for outcome 36
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese
Number analyzed (Participants) | 4 | 4 | 4 | 3
Ratio
  Day 5 | 1.250 (28) | 0.9972 (18) | 1.054 (9) | 1.022 (7)
  Day 10: number analyzed (Participants) | 4 | 3 | 4 | 3
  Day 10 | 1.163 (18) | 0.8962 (20) | 0.9605 (4) | 0.9412 (8)

38. Secondary Outcome: Part 2: Observed Accumulation Ratio for Cmax (Rac,Cmax) of PF-07817883 on Days 5 and 10
Description: Rac,Cmax of PF-07817883 was reported in this outcome measure. Rac,Cmax was calculated as Cmax on Day 5 or Day 10/Cmax on Day 1.
Time Frame: Day 5 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12 hours post-dose) and Day 10 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 hours post-dose)
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese
Number analyzed (Participants) | 4 | 4 | 4 | 3
Ratio
  Day 5 | 1.183 (22) | 1.075 (30) | 1.142 (33) | 0.9844 (18)
  Day 10: number analyzed (Participants) | 4 | 3 | 4 | 3
  Day 10 | 0.9744 (20) | 0.8471 (36) | 0.9717 (18) | 0.8712 (21)

39. Secondary Outcome: Part 2: Peak-to-Trough Ratio (PTR) of PF-07817883 on Days 5 and 10
Description: PTR of PF-07817883 was reported in this outcome measure. PTR was calculated as Cmax/Cmin.
Time Frame: as for outcome 38
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese
Number analyzed (Participants) | 4 | 4 | 4 | 3
Ratio
  Day 5 | 10.88 (10) | 13.47 (21) | 10.60 (49) | 13.22 (10)
  Day 10: number analyzed (Participants) | 4 | 3 | 4 | 3
  Day 10 | 8.566 (14) | 11.05 (30) | 10.13 (23) | 12.46 (9)

40. Secondary Outcome: Part 2: Apparent Clearance (CL/F) of PF-07817883 on Days 5 and 10
Description: CL/F of PF-07817883 was reported in this outcome measure. CL/F was calculated as dose/AUCinf.
Time Frame: as for outcome 38
Population: as for outcome 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour (L/hr)
Arm/Group | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese
Number analyzed (Participants) | 4 | 4 | 4 | 3
Liter/hour (L/hr)
  Day 5 | 10.83 (15) | 16.57 (10) | 13.12 (22) | 15.88 (29)
  Day 10: number analyzed (Participants) | 4 | 3 | 4 | 3
  Day 10 | 11.60 (10) | 17.13 (8) | 14.37 (18) | 17.32 (29)

41. Secondary Outcome: Part 2: Apparent Volume of Distribution (Vz/F) of PF-07817883 on Day 10
Description: Vz/F of PF-07817883 was reported in this outcome measure. Vz/F was calculated as dose/(AUCtau*kel).
Time Frame: Day 10 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 hours post-dose)
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese
Number analyzed (Participants) | 4 | 3 | 3 | 3
Liter | 200.1 (84) | 279.6 (62) | 198.1 (98) | 186.0 (115)

42. Secondary Outcome: Part 2: Terminal Half-Life (t1/2) of PF-07817883 on Day 10
Description: as for outcome 27
Time Frame: Day 10 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 hours post-dose)
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese
Number analyzed (Participants) | 4 | 3 | 3 | 3
Hours | 13.95 (9.3938) | 13.01 (8.8563) | 11.44 (6.8367) | 8.587 (5.8524)

43. Secondary Outcome: Part 2: Amount Excreted in Urine as Unchanged Drug Over the Dosing Interval Tau (Aetau) of PF-07817883 on Day 10
Description: Aetau was defined as amount excreted in urine as unchanged drug over the dosing interval tau, where tau= 12 hours. Aetau of PF-07817883 was reported in this outcome measure. Aetau was calculated as sum of (urine volume*urine concentration) for each collection over the dosing interval.
Time Frame: Day 10 (0 to 12 hours)
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligram (mg)
Arm/Group | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese
Number analyzed (Participants) | 4 | 3 | 4 | 3
Milligram (mg) | 18.47 (16) | 96.86 (5) | 373.2 (10) | 85.85 (20)

44. Secondary Outcome: Part 2: Percent of Dose Excreted in Urine as Unchanged Drug Over the Dosing Interval Tau (Aetau%) of PF-07817883 on Day 10
Description: Aetau% was defined as percentage of dose excreted in urine as unchanged drug over the dosing interval tau, where tau= 12 hours. Aetau% of PF-07817883 was reported in this outcome measure. Aetau% was calculated as 100*Aetau/dose.
Time Frame: Day 10 (0 to 12 hours)
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Percentage of Dose Excreted
Arm/Group | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese
Number analyzed (Participants) | 4 | 3 | 4 | 3
Percentage of Dose Excreted | 9.261 (16) | 16.15 (5) | 24.90 (10) | 14.34 (20)

45. Secondary Outcome: Part 2: Renal Clearance (CLr) of PF-07817883 on Day 10
Description: CLr of PF-07817883 was reported in this outcome measure. CLr was calculated as Aetau/AUCtau.
Time Frame: Day 10 (0 to 12 hours)
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour (L/hr)
Arm/Group | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese
Number analyzed (Participants) | 4 | 3 | 4 | 3
Liter/hour (L/hr) | 1.074 (20) | 2.771 (5) | 3.586 (26) | 2.477 (51)

46. Secondary Outcome: Part 3: Ratio Based on AUClast and AUCinf of Tablet Formulation Under Fed Condition and Fasted Condition
Description: Data for AUClast and AUCinf are reported in the descriptive section. AUClast was calculated by the linear/log trapezoidal method. AUCinf was calculated as AUClast + (Clast/kel), where Clast was the predicted plasma concentration at the last quantifiable time point from the log-linear regression analysis. Ratio based on AUClast and AUCinf of tablet formulations under fed and fasted conditions were reported in statistical analysis.
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 hours post-dose)
Population: Pharmacokinetic (PK) parameter set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of interest were reported. Here, ''Number Analyzed'' signifies participants evaluable for the specified rows. This outcome measure was planned to be analyzed only in the tablet formulation as pre-specified in the protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*Hour per milliliter (ng*hr/mL)
Arm/Group | Part 3: PF-07817883 SDD 600 mg (Tablet), Fasted | Part 3: PF-07817883 SDD 600 mg (Tablet), Fed | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fasted | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fed
Number analyzed (Participants) | 12 | 6 | 12 | 6
Nanogram*Hour per milliliter (ng*hr/mL)
  AUCinf: number analyzed (Participants) | 12 | 6 | 11 | 4
  AUCinf | 44140 (38) | 28430 (28) | 42930 (43) | 46170 (27)
  AUClast | 43570 (37) | 27750 (29) | 41620 (41) | 35930 (54)
Statistical Analysis 1: Comparison: Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fasted vs Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fed; AUCinf; Test type: Other; Ratio of Adjusted Geometric Means = 72.87, 90% CI 2-sided [60.98 to 87.09] — A paired t-test was used. Values had been back-transformed from natural log scale. Ratios (and 90% CIs) were expressed as percentages
Statistical Analysis 2: Comparison: Part 3: PF-07817883 SDD 600 mg (Tablet), Fasted vs Part 3: PF-07817883 SDD 600 mg (Tablet), Fed; AUCinf; Test type: Other; Ratio of Adjusted Geometric Means = 76.45, 90% CI 2-sided [68.35 to 85.52] — [estimate comment as in outcome 46, analysis 1]
Statistical Analysis 3: Comparison: Part 3: PF-07817883 SDD 600 mg (Tablet), Fasted vs Part 3: PF-07817883 SDD 600 mg (Tablet), Fed; AUClast; Test type: Other; Ratio of Adjusted Geometric Means = 73.52, 90% CI 2-sided [65.70 to 82.27] — [estimate comment as in outcome 46, analysis 1]
Statistical Analysis 4: Comparison: Part 3: PF-07817883 SDD 600 mg (Tablet), Fasted vs Part 3: PF-07817883 SDD 600 mg (Tablet), Fed; AUClast; Test type: Other; Ratio of Adjusted Geometric Means = 75.16, 90% CI 2-sided [66.36 to 85.13] — [estimate comment as in outcome 46, analysis 1]

47. Secondary Outcome: Part 3: Ratio Based on Maximum Observed Concentration (Cmax) of Tablet Formulation Under Fed Condition and Fasted Condition
Description: Data for Cmax are reported in the descriptive section. Ratio based on Cmax of tablet formulation under fed and fasted conditions were reported in statistical analysis.
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 hours post-dose)
Population: PK parameter set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of interest were reported. This outcome measure was planned to be analyzed only in the tablet formulation as pre-specified in the protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | Part 3: PF-07817883 SDD 600 mg (Tablet), Fasted | Part 3: PF-07817883 SDD 600 mg (Tablet), Fed | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fasted | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fed
Number analyzed (Participants) | 12 | 6 | 12 | 6
Nanogram per milliliter (ng/mL) | 6934 (35) | 4590 (21) | 6284 (38) | 5008 (47)
Statistical Analysis 1: Comparison: Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fasted vs Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fed; Test type: Other; Ratio of Adjusted Geometric Means = 76.72, 90% CI 2-sided [60.21 to 97.75] — [estimate comment as in outcome 46, analysis 1]
Statistical Analysis 2: Comparison: Part 3: PF-07817883 SDD 600 mg (Tablet), Fasted vs Part 3: PF-07817883 SDD 600 mg (Tablet), Fed; Test type: Other; Ratio of Adjusted Geometric Means = 70.92, 90% CI 2-sided [53.70 to 93.67] — [estimate comment as in outcome 46, analysis 1]

48. Secondary Outcome: Part 3: Time for Cmax (Tmax) of PF-07817883
Description: Tmax of PF-07817883 was reported in this outcome measure.
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 hours post-dose)
Population: Pharmacokinetic (PK) parameter set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of interest were reported.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 3: PF-07817883 600 mg (Suspension), Fasted | Part 3: PF-07817883 SDD 600 mg (Tablet), Fasted | Part 3: PF-07817883 SDD 600 mg (Tablet), Fed | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fasted | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fed
Number analyzed (Participants) | 12 | 12 | 6 | 12 | 6
Hours | 0.750 [0.500 to 1.05] | 1.01 [0.500 to 2.00] | 4.00 [1.00 to 4.00] | 1.34 [1.00 to 2.00] | 4.00 [2.00 to 6.00]

49. Secondary Outcome: Part 3: Maximum Observed Concentration (Cmax) of PF-07817883
Description: Cmax of PF-07817883 was reported in this outcome measure.
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 hours post-dose)
Population: as for outcome 48
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter (ng/mL)
Arm/Group | Part 3: PF-07817883 600 mg (Suspension), Fasted | Part 3: PF-07817883 SDD 600 mg (Tablet), Fasted | Part 3: PF-07817883 SDD 600 mg (Tablet), Fed | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fasted | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fed
Number analyzed (Participants) | 12 | 12 | 6 | 12 | 6
Nanogram/milliliter (ng/mL) | 9354 (18) | 6934 (35) | 4590 (21) | 6284 (38) | 5008 (47)

50. Secondary Outcome: Part 3: Area Under Plasma Concentration Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of PF-07817883
Description: as for outcome 22
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 hours post-dose)
Population: as for outcome 48
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | Part 3: PF-07817883 600 mg (Suspension), Fasted | Part 3: PF-07817883 SDD 600 mg (Tablet), Fasted | Part 3: PF-07817883 SDD 600 mg (Tablet), Fed | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fasted | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fed
Number analyzed (Participants) | 12 | 12 | 6 | 12 | 6
Nanogram*hour/milliliter (ng*hr/mL) | 42540 (35) | 43570 (37) | 27750 (29) | 41620 (41) | 35930 (54)

51. Secondary Outcome: Part 3: Area Under the Concentration -Time Curve From Time Zero (0) Extrapolated to Infinite Time (AUCinf) of PF-07817883
Description: as for outcome 25
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 hours post-dose)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | Part 3: PF-07817883 600 mg (Suspension), Fasted | Part 3: PF-07817883 SDD 600 mg (Tablet), Fasted | Part 3: PF-07817883 SDD 600 mg (Tablet), Fed | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fasted | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fed
Number analyzed (Participants) | 12 | 12 | 6 | 11 | 4
Nanogram*hour/milliliter (ng*hr/mL) | 42970 (35) | 44140 (38) | 28430 (28) | 42930 (43) | 46170 (27)

52. Secondary Outcome: Part 3: Terminal Half-Life (t1/2) of PF-07817883
Description: as for outcome 27
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 hours post-dose)
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part 3: PF-07817883 600 mg (Suspension), Fasted | Part 3: PF-07817883 SDD 600 mg (Tablet), Fasted | Part 3: PF-07817883 SDD 600 mg (Tablet), Fed | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fasted | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fed
Number analyzed (Participants) | 12 | 12 | 6 | 11 | 4
Hours | 7.578 (3.2536) | 7.957 (3.8740) | 10.15 (2.2890) | 6.822 (3.5964) | 11.07 (4.4518)

53. Secondary Outcome: Part 3: Apparent Clearance (CL/F) of PF-07817883
Description: CL/F of PF-07817883 was reported in this outcome measure. CL/F was calculated as dose/AUCinf.
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 hours post-dose)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour
Arm/Group | Part 3: PF-07817883 600 mg (Suspension), Fasted | Part 3: PF-07817883 SDD 600 mg (Tablet), Fasted | Part 3: PF-07817883 SDD 600 mg (Tablet), Fed | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fasted | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fed
Number analyzed (Participants) | 12 | 12 | 6 | 11 | 4
Liter/hour | 13.97 (35) | 13.58 (38) | 21.09 (28) | 13.98 (43) | 12.98 (27)

54. Secondary Outcome: Part 3: Apparent Volume of Distribution (Vz/F) of PF-07817883
Description: Vz/F of PF-07817883 was reported in this outcome measure. Vz/F was calculated as dose/(AUCtau*kel).
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48 hours post-dose)
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Part 3: PF-07817883 600 mg (Suspension), Fasted | Part 3: PF-07817883 SDD 600 mg (Tablet), Fasted | Part 3: PF-07817883 SDD 600 mg (Tablet), Fed | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fasted | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fed
Number analyzed (Participants) | 12 | 12 | 6 | 11 | 4
Liter | 136.2 (55) | 136.7 (50) | 302.2 (31) | 120.7 (55) | 192.8 (64)

55. Secondary Outcome: Part 3: Number of Participants With TEAEs
Description: as for outcome 5
Time Frame: From start of study treatment up to 29-36 days after administration of last dose of study intervention (maximum up to 49 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3: PF-07817883 600 mg (Suspension), Fasted | Part 3: PF-07817883 SDD 600 mg (Tablet), Fasted | Part 3: PF-07817883 SDD 600 mg (Tablet), Fed | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fasted | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fed
Number analyzed (Participants) | 12 | 12 | 6 | 12 | 6
Participants | 4 | 1 | 1 | 4 | 2

56. Secondary Outcome: Part 3: Number of Participants With Laboratory Test Abnormalities
Description: Laboratory parameters included: hematology (monocytes/leukocytes >1.2*ULN [%], partial thromboplastin time >1.1*ULN [seconds]) and urinalysis (urine hemoglobin >=1, bacteria >20 [/lpf]). Number of participants with any lab test abnormalities meeting the pre-specified criteria are reported in this outcome measure.
Time Frame: as for outcome 55
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3: PF-07817883 600 mg (Suspension), Fasted | Part 3: PF-07817883 SDD 600 mg (Tablet), Fasted | Part 3: PF-07817883 SDD 600 mg (Tablet), Fed | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fasted | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fed
Number analyzed (Participants) | 12 | 12 | 6 | 2 | 6
Participants | 0 | 0 | 2 | 0 | 2

57. Secondary Outcome: Part 3: Number of Participants With Vital Signs Meeting Pre-Defined Criteria
Description: as for outcome 7
Time Frame: Up to Day 3 of each period
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Part 3: PF-07817883 600 mg (Suspension), Fasted: Participants received PF-07817883 600 mg oral suspension under fasted conditions. An overnight fast for approximately 10 hours was required.
- Part 3: PF-07817883 SDD 600 mg (Tablet), Fasted: Participants received PF-07817883 600 mg spray dried dispersion (SDD) under fasted conditions. An overnight fast for approximately 10 hours was required. Participants swallowed PF-07817883 as whole and did not chew prior to swallowing.
- Part 3: PF-07817883 SDD 600 mg (Tablet), Fed: Participants received PF-07817883 600 mg spray dried dispersion (SDD) under fed conditions. PF-07817883 was administered approximately 10 minutes after finishing the meal/snack. Participants swallowed PF-07817883 as whole and did not chew prior to swallowing.
- Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fasted: Participants received PF-07817883 600 mg crystalline tablet under fasted conditions. An overnight fast for approximately 10 hours was required. Participants swallowed PF-07817883 as whole and did not chew prior to swallowing.
- Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fed: Participants received PF-07817883 600 mg crystalline tablet under fed conditions. PF-07817883 was administered approximately 10 minutes after finishing the meal/snack. Participants swallowed PF-07817883 as whole and did not chew prior to swallowing.
Arm/Group | Part 3: PF-07817883 600 mg (Suspension), Fasted | Part 3: PF-07817883 SDD 600 mg (Tablet), Fasted | Part 3: PF-07817883 SDD 600 mg (Tablet), Fed | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fasted | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fed
Number analyzed (Participants) | 12 | 12 | 6 | 12 | 6
Participants | 0 | 0 | 0 | 0 | 0

58. Secondary Outcome: Part 3: Number of Participants With ECG Abnormalities
Description: as for outcome 4
Time Frame: Up to Day 3 of each period
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3: PF-07817883 600 mg (Suspension), Fasted | Part 3: PF-07817883 SDD 600 mg (Tablet), Fasted | Part 3: PF-07817883 SDD 600 mg (Tablet), Fed | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fasted | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fed
Number analyzed (Participants) | 12 | 12 | 6 | 12 | 6
Participants | 0 | 0 | 0 | 0 | 0

59. Secondary Outcome: Part 4: Time for Cmax (Tmax) of PF-07817883
Description: Tmax of PF-07817883 was reported in this outcome measure.
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48, 72 hours post-dose)
Population: as for outcome 10
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 4: PF-07817883 600 mg (Suspension), Fasted
Number analyzed (Participants) | 6
Hours | 0.500 [0.500 to 2.00]

60. Secondary Outcome: Part 4: Maximum Observed Concentration (Cmax) of PF-07817883
Description: Cmax of PF-07817883 was reported in this outcome measure.
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48, 72 hours post-dose)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter (ng/mL)
Arm/Group | Part 4: PF-07817883 600 mg (Suspension), Fasted
Number analyzed (Participants) | 6
Nanogram/milliliter (ng/mL) | 6791 (35)

61. Secondary Outcome: Part 4: Area Under Plasma Concentration Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of PF-07817883
Description: as for outcome 22
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48, 72 hours post-dose)
Population: as for outcome 10
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | Part 4: PF-07817883 600 mg (Suspension), Fasted
Number analyzed (Participants) | 6
Nanogram*hour/milliliter (ng*hr/mL) | 35520 (24)

62. Secondary Outcome: Part 4: Area Under the Concentration -Time Curve From Time Zero (0) Extrapolated to Infinite Time (AUCinf) of PF-07817883
Description: as for outcome 25
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48, 72 hours post-dose)
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | Part 4: PF-07817883 600 mg (Suspension), Fasted
Number analyzed (Participants) | 5
Nanogram*hour/milliliter (ng*hr/mL) | 36910 (26)

63. Secondary Outcome: Part 4: Terminal Half-Life (t1/2) of PF-07817883
Description: as for outcome 27
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48, 72 hours post-dose)
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Part 4: PF-07817883 600 mg (Suspension), Fasted
Number analyzed (Participants) | 5
Hours | 6.882 (3.0621)

64. Secondary Outcome: Part 4: Apparent Clearance (CL/F) of PF-07817883
Description: CL/F of PF-07817883 was reported in this outcome measure. CL/F was calculated as dose/AUCinf.
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48, 72 hours post-dose)
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour
Arm/Group | Part 4: PF-07817883 600 mg (Suspension), Fasted
Number analyzed (Participants) | 5
Liter/hour | 16.26 (26)

65. Secondary Outcome: Part 4: Apparent Volume of Distribution (Vz/F) of PF-07817883
Description: Vz/F of PF-07817883 was reported in this outcome measure. Vz/F was calculated as dose/(AUCtau*kel).
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 4, 6, 8, 12, 16, 24, 48, 72 hours post-dose)
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | Part 4: PF-07817883 600 mg (Suspension), Fasted
Number analyzed (Participants) | 5
Liter | 146.7 (36)

66. Secondary Outcome: Part 4: Number of Participants With TEAEs
Description: as for outcome 5
Time Frame: From start of study treatment up to 29-36 days after administration of last dose of study intervention (maximum up to 47 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 4: PF-07817883 600 mg (Suspension), Fasted
Number analyzed (Participants) | 6
Participants | 4

67. Secondary Outcome: Part 4: Number of Participants With Laboratory Test Abnormalities
Description: Laboratory parameters included: hematology (mean corpuscular volume <0.9*LLN [cubic micrometer {um^3}], mean corpuscular hemoglobin <0.9*LLN [picograms per cell {pg/cell}], monocytes/leukocytes >1.2*ULN [%]). Number of participants with any lab test abnormalities meeting the pre-specified criteria are reported in this outcome measure.
Time Frame: as for outcome 66
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 4: PF-07817883 600 mg (Suspension), Fasted
Number analyzed (Participants) | 6
Participants | 1

68. Secondary Outcome: Part 4: Number of Participants With Vital Signs Meeting Pre-Defined Criteria
Description: as for outcome 18
Time Frame: Up to Day 11
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 4: PF-07817883 600 mg (Suspension), Fasted
Number analyzed (Participants) | 6
Participants
  SBP value < 90 mmHg | 1
  SBP change >= 30 mmHg increase | 0
  SBP change >= 30 mmHg decrease | 0
  DBP value < 50 mmHg | 1
  DBP change >= 20 mmHg increase | 0
  DBP change >= 20 mmHg decrease | 0
  Pulse rate value < 40 bpm | 0
  Pulse rate value > 120 bpm | 0

69. Secondary Outcome: Part 4: Number of Participants With ECG Abnormalities
Description: as for outcome 4
Time Frame: Up to Day 11
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Part 4: PF-07817883 600 mg (Suspension), Fasted
Number analyzed (Participants) | 6
Participants | 0

70. Secondary Outcome: Part 5: Number of Participants With TEAEs
Description: as for outcome 5
Time Frame: From start of study treatment up to 38-45 days after administration of last dose of study intervention (maximum up to 65 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07817883 600 mg (Suspension) BID/ Midazolam 5 mg | Midazolam 5 mg
Number analyzed (Participants) | 13 | 13
Participants | 11 | 10

71. Secondary Outcome: Part 5: Number of Participants With Laboratory Test Abnormalities
Description: Laboratory parameters included: hematology (lymphocytes <0.8*LLN [10^3/mm3], lymphocytes/leukocytes <0.8*LLN [%], neutrophils/leukocytes <0.8*LLN [%], monocytes/leukocytes >1.2*ULN [%]), chemistry (amylase >1.5*ULN [units/liter] {U/L}), and urinalysis (urine hemoglobin >=1). Number of participants with any lab test abnormalities meeting the pre-specified criteria are reported in this outcome measure.
Time Frame: as for outcome 70
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07817883 600 mg (Suspension) BID/ Midazolam 5 mg | Midazolam 5 mg
Number analyzed (Participants) | 13 | 7
Participants | 5 | 2

72. Secondary Outcome: Part 5: Number of Participants With Vital Signs Meeting Pre-Defined Criteria
Description: as for outcome 18
Time Frame: as for outcome 70
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07817883 600 mg (Suspension) BID/ Midazolam 5 mg | Midazolam 5 mg
Number analyzed (Participants) | 13 | 13
Participants
  SBP value < 90 mmHg | 3 | 3
  SBP change >= 30 mmHg increase | 0 | 0
  SBP change >= 30 mmHg decrease | 0 | 1
  DBP value < 50 mmHg | 2 | 2
  DBP change >= 20 mmHg increase | 0 | 0
  DBP change >= 20 mmHg decrease | 0 | 0
  Pulse rate value < 40 bpm | 0 | 0
  Pulse rate value > 120 bpm | 0 | 0

73. Secondary Outcome: Part 5: Number of Participants With ECG Abnormalities
Description: as for outcome 4
Time Frame: as for outcome 70
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PF-07817883 600 mg (Suspension) BID/ Midazolam 5 mg | Midazolam 5 mg
Number analyzed (Participants) | 13 | 13
Participants | 0 | 0

74. Secondary Outcome: Part 5: Time for Cmax (Tmax) of Midazolam
Description: Tmax of midazolam was reported in this outcome measure.
Time Frame: as for outcome 14
Population: as for outcome 25
Measure: Median (Full Range); unit: Hours
Arm/Group | PF-07817883 600 mg (Suspension) BID/ Midazolam 5 mg | Midazolam 5 mg
Number analyzed (Participants) | 12 | 13
Hours | 0.500 [0.500 to 1.12] | 0.500 [0.500 to 1.02]

75. Secondary Outcome: Part 5: Area Under Plasma Concentration Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of Midazolam
Description: AUClast of midazolam was reported in this outcome measure. AUClast was calculated by the linear/log trapezoidal method.
Time Frame: as for outcome 14
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | PF-07817883 600 mg (Suspension) BID/ Midazolam 5 mg | Midazolam 5 mg
Number analyzed (Participants) | 12 | 13
Nanogram*hour/milliliter (ng*hr/mL) | 92.37 (27) | 77.46 (32)

76. Secondary Outcome: Part 5: Terminal Half-Life (t1/2) of Midazolam
Description: t1/2 of midazolam was reported in this outcome measure. t1/2 was calculated by Loge(2)/kel, where kel was the terminal phase rate constant calculated by a linear regression of the log linear concentration-time curve. Only those data points judged to describe the terminal log-linear decline were used in the regression.
Time Frame: as for outcome 14
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | PF-07817883 600 mg (Suspension) BID/ Midazolam 5 mg | Midazolam 5 mg
Number analyzed (Participants) | 12 | 13
Hours | 6.589 (1.6566) | 6.923 (1.9185)

77. Secondary Outcome: Part 5: Apparent Clearance (CL/F) of Midazolam
Description: CL/F of midazolam was reported in this outcome measure. CL/F was calculated as dose/AUCinf.
Time Frame: as for outcome 14
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter/hour
Arm/Group | PF-07817883 600 mg (Suspension) BID/ Midazolam 5 mg | Midazolam 5 mg
Number analyzed (Participants) | 12 | 13
Liter/hour | 53.02 (26) | 62.60 (31)

78. Secondary Outcome: Part 5: Apparent Volume of Distribution (Vz/F) of Midazolam
Description: Vz/F of midazolam was reported in this outcome measure. Vz/F was calculated as dose/(AUCinf*kel).
Time Frame: as for outcome 14
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liter
Arm/Group | PF-07817883 600 mg (Suspension) BID/ Midazolam 5 mg | Midazolam 5 mg
Number analyzed (Participants) | 12 | 13
Liter | 488.5 (44) | 598.9 (45)

79. Secondary Outcome: Part 6: Maximum Observed Concentration (Cmax) of PF-07817883
Description: Cmax of PF-07817883 was reported in this outcome measure.
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose)
Population: PK parameter set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of interest were reported. This outcome measure was planned to be analyzed only in the PF-07817883 6000 mg (suspension), fasted arm, as pre-specified in the protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram/milliliter (ng/mL)
Arm/Group | PF-07817883 6000 mg (Suspension), Fasted
Number analyzed (Participants) | 23
Nanogram/milliliter (ng/mL) | 53160 (21)

80. Secondary Outcome: Part 6: Time for Cmax (Tmax) of PF-07817883
Description: Tmax of PF-07817883 was reported in this outcome measure.
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose)
Population: as for outcome 79
Measure: Median (Full Range); unit: Hours
Arm/Group | PF-07817883 6000 mg (Suspension), Fasted
Number analyzed (Participants) | 23
Hours | 1.00 [0.567 to 1.50]

81. Secondary Outcome: Part 6: Area Under Plasma Concentration Time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUClast) of PF-07817883
Description: as for outcome 22
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose)
Population: as for outcome 79
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | PF-07817883 6000 mg (Suspension), Fasted
Number analyzed (Participants) | 23
Nanogram*hour/milliliter (ng*hr/mL) | 248300 (17)

82. Secondary Outcome: Part 6: Area Under the Concentration -Time Curve From Time Zero (0) Extrapolated to Infinite Time (AUCinf) of PF-07817883
Description: as for outcome 25
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose)
Population: PK parameter set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention and in whom at least 1 of the PK parameters of interest were reported. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure. This outcome measure was planned to be analyzed only in the PF-07817883 6000 mg (suspension), fasted arm, as pre-specified in the protocol.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanogram*hour/milliliter (ng*hr/mL)
Arm/Group | PF-07817883 6000 mg (Suspension), Fasted
Number analyzed (Participants) | 19
Nanogram*hour/milliliter (ng*hr/mL) | 253000 (17)

83. Secondary Outcome: Part 6: Terminal Half-Life (t1/2) of PF-07817883
Description: as for outcome 27
Time Frame: Day 1 (pre-dose, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose)
Population: as for outcome 82
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | PF-07817883 6000 mg (Suspension), Fasted
Number analyzed (Participants) | 19
Hours | 12.64 (7.1787)

ADVERSE EVENTS:
Time Frame: Part 1 and Part 6: From start of study treatment up to 28-35 days after administration of last dose of study intervention (maximum up to 48 and 52 days respectively); Part 2 and Part 5: From start of study treatment up to 38-45 days after administration of last dose of study intervention (maximum up to 55 and 65 days respectively); Part 3 and Part 4: From start of study treatment up to 29-36 days after administration of last dose of study intervention (maximum up to 49 and 47 days respectively)
Description: Safety population included all participants randomly assigned to study intervention, who took at least 1 dose of study intervention. Participants were analyzed according to the product they actually received.
Groups:
- Part 1: Placebo (Suspension), Fasted: Participants who received a single dose of placebo as an oral suspension on Day 1 of either Period 1, 2 or 3 under fasted conditions were included.
- Part 1: Placebo (Suspension), Fed: Participants who received a single dose of placebo as an oral suspension on Day 1 of either Period 1, 2 or 3 under fed conditions were included.
- Part 1: PF-07817883 150 mg (Suspension), Fasted: Participants who received a single dose of PF-07817883 150 mg as an oral suspension on Day 1 of either Period 1, 2 or 3 under fasted conditions were included.
- Part 1: PF-07817883 500 mg (Suspension), Fasted: Participants who received a single dose of PF-07817883 500 mg as an oral suspension on Day 1 of either Period 1, 2 or 3 under fasted conditions were included.
- Part 1: PF-07817883 500 mg (Suspension), Fed: Participants who received a single dose of PF-07817883 500 mg as an oral suspension on Day 1 of either Period 1, 2 or 3 under fed conditions were included.
- Part 1: PF-07817883 1500 mg (Suspension), Fasted: Participants who received a single dose of PF-07817883 1500 mg as an oral suspension on Day 1 of either Period 1, 2 or 3 under fasted conditions were included.
- Part 1: PF-07817883 3000 mg (Suspension), Fasted: Participants who received a single dose of PF-07817883 3000 mg as an oral suspension on Day 1 of either Period 1, 2 or 3 under fasted conditions were included.
- Part 1: PF-07817883 4000 mg (Suspension), Fasted: Participants who received a single dose of PF-07817883 4000 mg as an oral suspension on Day 1 of either Period 1, 2 or 3 under fasted conditions were included.
- Part 5: PF-07817883 600 mg (Suspension) BID/ Midazolam 5 mg: Participants received PF-07817883 600 mg oral suspension twice a day (BID) for 10 days (Day 1 morning to Day 10 morning). On Day 10 morning, participants received a single oral dose of 5 mg midazolam administered with PF-07817883.
- Part 5: Midazolam 5 mg: Participants received oral solution of Midazolam 5 mg on Day 1 of either Period 1 or 2.
- Part 6: Placebo (Suspension), Fasted: Participants received Placebo oral suspension at 0 and 1 hours on Day 1 of either Period 1, 2 or 3 following an overnight fast of at least 10 hours.
- Part 6: PF-07817883 6000 mg (Suspension), Fasted: Participants received 6000 mg PF-07817883 oral suspension administered as two split doses of 3000 mg at 0 and 1 hour on Day 1 of either Period 1, 2 or 3 following an overnight fast of at least 10 hours.
- Part 6: Moxifloxacin 400 mg, Fasted: Participants received 400 mg Moxifloxacin oral tablet and placebo at 0 and 1 hour respectively on Day 1 of either Period 1, 2 or 3 following an overnight fast of at least 10 hours.
Arm/Group | Part 1: Placebo (Suspension), Fasted | Part 1: Placebo (Suspension), Fed | Part 1: PF-07817883 150 mg (Suspension), Fasted | Part 1: PF-07817883 500 mg (Suspension), Fasted | Part 1: PF-07817883 500 mg (Suspension), Fed | Part 1: PF-07817883 1500 mg (Suspension), Fasted | Part 1: PF-07817883 3000 mg (Suspension), Fasted | Part 1: PF-07817883 4000 mg (Suspension), Fasted | Part 2: Placebo (Suspension) BID, Fasted | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted | Part 2: Placebo (Suspension) BID, Fasted, Chinese | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese | Part 3: PF-07817883 600 mg (Suspension), Fasted | Part 3: PF-07817883 SDD 600 mg (Tablet), Fasted | Part 3: PF-07817883 SDD 600 mg (Tablet), Fed | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fasted | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fed | Part 4: PF-07817883 600 mg (Suspension), Fasted | Part 5: PF-07817883 600 mg (Suspension) BID/ Midazolam 5 mg | Part 5: Midazolam 5 mg | Part 6: Placebo (Suspension), Fasted | Part 6: PF-07817883 6000 mg (Suspension), Fasted | Part 6: Moxifloxacin 400 mg, Fasted
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/2 | 0/6 | 0/6 | 0/4 | 0/6 | 0/5 | 0/5 | 0/6 | 0/4 | 0/4 | 0/4 | 0/1 | 0/3 | 0/12 | 0/12 | 0/6 | 0/12 | 0/6 | 0/6 | 0/13 | 0/13 | 0/23 | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/2 | 0/6 | 0/6 | 0/4 | 0/6 | 0/5 | 0/5 | 0/6 | 0/4 | 0/4 | 0/4 | 0/1 | 0/3 | 0/12 | 0/12 | 0/6 | 0/12 | 0/6 | 0/6 | 0/13 | 0/13 | 0/23 | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 4/10 | 1/2 | 2/6 | 1/6 | 0/4 | 3/6 | 0/5 | 1/5 | 2/6 | 1/4 | 0/4 | 2/4 | 0/1 | 2/3 | 4/12 | 1/12 | 1/6 | 4/12 | 2/6 | 4/6 | 11/13 | 10/13 | 0/23 | 0/23 | 0/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Placebo (Suspension), Fasted (N=10) | Part 1: Placebo (Suspension), Fed (N=2) | Part 1: PF-07817883 150 mg (Suspension), Fasted (N=6) | Part 1: PF-07817883 500 mg (Suspension), Fasted (N=6) | Part 1: PF-07817883 500 mg (Suspension), Fed (N=4) | Part 1: PF-07817883 1500 mg (Suspension), Fasted (N=6) | Part 1: PF-07817883 3000 mg (Suspension), Fasted (N=5) | Part 1: PF-07817883 4000 mg (Suspension), Fasted (N=5) | Part 2: Placebo (Suspension) BID, Fasted (N=6) | Part 2: PF-07817883 200 mg (Suspension) BID, Fasted (N=4) | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted (N=4) | Part 2: PF-07817883 1500 mg (Suspension) BID, Fasted (N=4) | Part 2: Placebo (Suspension) BID, Fasted, Chinese (N=1) | Part 2: PF-07817883 600 mg (Suspension) BID, Fasted, Chinese (N=3) | Part 3: PF-07817883 600 mg (Suspension), Fasted (N=12) | Part 3: PF-07817883 SDD 600 mg (Tablet), Fasted (N=12) | Part 3: PF-07817883 SDD 600 mg (Tablet), Fed (N=6) | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fasted (N=12) | Part 3: PF-07817883 Crystalline 600 mg (Tablet), Fed (N=6) | Part 4: PF-07817883 600 mg (Suspension), Fasted (N=6) | Part 5: PF-07817883 600 mg (Suspension) BID/ Midazolam 5 mg (N=13) | Part 5: Midazolam 5 mg (N=13) | Part 6: Placebo (Suspension), Fasted (N=23) | Part 6: PF-07817883 6000 mg (Suspension), Fasted (N=23) | Part 6: Moxifloxacin 400 mg, Fasted (N=24)
Constipation (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urine output decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Defaecation urgency (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vessel puncture site bruise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pseudofolliculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urine output increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 9 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-03-09): https://cdn.clinicaltrials.gov/large-docs/03/NCT05580003/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-24): https://cdn.clinicaltrials.gov/large-docs/03/NCT05580003/SAP_001.pdf